

## STATISTICAL ANALYSIS PLAN

Protocol title: A randomized, double blind, placebo-controlled,

multi-center, parallel group study to evaluate the efficacy and safety of dupilumab in patients with prurigo nodularis who are inadequately controlled on

topical prescription therapies or when those

therapies are not advisable

Protocol number: EFC16460

Compound number SAR231893/REGN668 (INN/Trademark): dupilumab/Dupixent

Study phase: Phase 3

Short title: Study of dupilumab for the treatment of patients with

prurigo nodularis, inadequately controlled on topical prescription therapies or when those therapies are

not advisable

**LIBERTY-PN PRIME 2** 

Statistician:

Statistical project leader:

Date of issue: 08-Aug-2021

Regulatory agency identifier number(s):

IND: IND107969

EudraCT: 2019-003801-90
NCT: NCT04202679
WHO: U1111-1241-8174

Other: Not applicable

Total number of pages: 64

Any and all information presented in this document shall be treated as confidential and shall remain the exclusive property of Sanofi (or any of its affiliated companies). The use of such confidential information must be restricted to the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated to any unauthorized persons, for any reason, in any form whatsoever without the prior written consent of Sanofi (or the concerned affiliated company); 'affiliated company' means any corporation, partnership or other entity which at the date of communication or afterwards (i) controls directly or indirectly Sanofi, (ii) is directly or indirectly controlled by Sanofi, with 'control' meaning direct or indirect ownership of more than 50% of the capital stock or the voting rights in such corporation, partnership or other entity

According to template: QSD-002643 VERSION 8.0 (17-JUN-2020)

## **TABLE OF CONTENTS**

| STATIS | STICAL ANALYSIS PLAN | 1 |
|---------|-------------------------------------------|----|
| TABLE | OF CONTENTS | 2 |
| LIST O | F TABLES | |
| | ON HISTORY | |
| 1 | INTRODUCTION | 7 |
| 1.1 | STUDY DESIGN | 7 |
| 1.2 | OBJECTIVE AND ENDPOINTS | 7 |
| 1.2.1 | Estimands | 10 |
| 2 | SAMPLE SIZE DETERMINATION | 14 |
| 3 | ANALYSIS POPULATIONS | 15 |
| 4 | STATISTICAL ANALYSES | 17 |
| 4.1 | GENERAL CONSIDERATIONS | 17 |
| 4.2 | PARTICIPANT DISPOSITIONS | 17 |
| 4.3 | PRIMARY ENDPOINT(S) ANALYSIS | 18 |
| 4.3.1 | Definition of endpoint(s) | 18 |
| 4.3.2 | Main analytical approach | 20 |
| 4.3.3 | Sensitivity analysis | |
| 4.3.4 | Supplementary analyses | 21 |
| 4.3.5 | Subgroup analyses | 22 |
| 4.4 | SECONDARY ENDPOINT(S) ANALYSIS | 23 |
| 4.4.1 | Key/Confirmatory secondary endpoint(s) | 23 |
| 4.4.1.1 | ······ -·· (- / ········ | |
| 4.4.1.2 | 7 11 | |
| 4.4.2 | Supportive secondary endpoint(s) | 24 |
| 4.5 | TERTIARY/EXPLORATORY ENDPOINT(S) ANALYSIS | 26 |
| 4.5.1 | Definition of endpoint(s) | 26 |
| 4.5.2 | Main analytical approach | 29 |
| 4.6 | MULTIPLICITY ISSUES | 29 |

| 4.7 | SAFETY ANALYSES | 30 |
|---|---|---|
| 4.7.1 | Extent of exposure | 30 |
| 4.7.2 | Adverse events | 31 |
| 4.7.3 | Additional safety assessments | |
| 4.7.3.1 | Laboratory variables, vital signs and electrocardiograms (ECGs) | 36 |
| 4.8 | OTHER ANALYSES | 38 |
| 4.8.1 | Pharmacokinetic analyses | 38 |
| 4.8.2 | Immunogenicity analyses | 39 |
| 4.8.3 | Pharmacodynamic/genomics endpoints | 41 |
| 4.9 | INTERIM ANALYSES | 42 |
| 5 | SUPPORTING DOCUMENTATION | 43 |
| 5.1 | APPENDIX 1 LIST OF ABBREVIATIONS | 43 |
| 5.2 | APPENDIX 2 CHANGES TO PROTOCOL-PLANNED ANALYSES | 45 |
| 5.3 | APPENDIX 3 DEMOGRAPHICS AND BASELINE CHARACTERISTICS, PRIOR OR CONCOMITANT MEDICATIONS/PROCEDURES | 46 |
| 5.4 | APPENDIX 4 DATA HANDLING CONVENTIONS | 50 |
| 5.5 | APPENDIX 5 SAMPLE SAS CODE | 57 |
| 5.6 | APPENDIX 6 SELECTION CRITERIA FOR AE/MEDICATION GROUPINGS | 59 |
| 5.7 | APPENDIX 7 MEDICATION/PROCEDURE ADJUDICATION ALGORITHM | 61 |
| 6 | DEEEDENCES | 6/ |

## **LIST OF TABLES**

| Fable 1 - Major changes in statistical analysis plan | 5 |
|---|---|
| Гable 2 - Objectives and endpoints | 7 |
| Fable 3 - Summary of primary estimand for main endpoints | 11 |
| Гable 4 - Populations for analyses | 15 |
| Table 5 - Prohibited medications/procedures and rescue medications that impact efficacy | 19 |
| Гable 6 - Sorting of AE tables | 32 |
| Table 7 - Analyses of adverse events | 33 |
| Γable 8 - Selections for AESIs and other AEs of interest | 34 |
| Table 9 - Major statistical changes in protocol amendment(s) | 45 |
| Table 10 - Time window for eDiary efficacy variables | 51 |
| Table 11 - Time window for efficacy variables | 53 |
| Table 12 - Time window for safety endpoints | 55 |
| Fable 13 - Time window for pharmacokinetics/pharmacodynamics variables | 56 |
| Table 1/1 - List of PTs or Medications for CMOs/CDGs | 50 |

## **VERSION HISTORY**

This Statistical Analysis Plan (SAP) for study EFC16460 is based on the Protocol Amendment 1 dated 20-May-2020 and a health authority's feedback on EFC16459 Protocol Amendment 2 dated 14-Apr-2021 (See EFC16459 SAP for details). This section summarizes major changes to the statistical analysis features in the SAP. All changes to the statistical analysis features from the original protocol to Amendment 1 are described in Appendix 2.

Table 1 - Major changes in statistical analysis plan

| SAP<br>Version | Approval<br>Date | Changes | Rationale |
|---|---|---|---|
| 1.0 | 04-Feb-2021 | Not Applicable | Original version |
| 2.0 | Current version | Add objective "To demonstrate efficacy of dupilumab on both itch as well as skin lesions within the same participant" and multicomponent endpoint (Proportion of participants with both an improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24 and an IGA PN-S 0 or 1 score at Week 24) as a key secondary endpoint for the US and US reference countries hierarchy. | To add this multicomponent endpoint as another measure of treatment success based on feedback from a health authority. |
| | | Add supplementary analysis (tipping point analyses) for primary and key secondary endpoints | This additional supplementary analysis was recommended by a health authority to assess whether the estimate, and the inference thereof, was robust to departure from the strategies used in primary analysis for handling intercurrent events and missing data. |
| | | Add subgroup analyses for key secondary endpoints. | To evaluate whether the treatment effect is consistent across pre-specified subgroups on the key secondary endpoints in addition to the primary endpoint. |
| | | Add subgroup analyses for participants who have been impacted (or not) by COVID-19 | To address a health authority's request to assess the impact of the treatment effect by COVID-19. |
| | | Modify hierarchical order for multiplicity procedure for US and US reference countries | To include the multicomponent endpoint in the hierarchy to address the health authority's feedback requesting assessment of this endpoint as another measure of treatment success. |
| | | Add as-observed plus multiple imputation supplementary analysis for the secondary endpoint (percent change from baseline in WI-NRS at Week 24) | To explore the robustness of the estimate, and the inference thereof, with a different strategy for handling intercurrent events and missing data |
| | | Remove "selected" in the text including "selected prohibited and/or rescue medication" | Since a participant who takes any protocol specified prohibited medications/procedures and/or rescue |

| SAP<br>Version | Approval<br>Date | Changes | Rationale |
|---|---|---|---|
| | | | medications is considered as a non-<br>responder after medical<br>adjudication/confirmation conducted in a<br>blinded fashion, use of the word<br>"selected" is confusing. |
| | | Add additional exposure-adjusted adverse event incidence rate tables that will provide the number of patients with at least 1 event per 100 patient-years. | As requested by a health authority to include exposure-adjusted incidence rate and patient years in the summaries for TEAEs and AESIs. |
| | | Added "Keratitis FDA" to other AE groupings | For consistency with other dupilumab studies |

The first participant was randomized on 2020-02-03.

## 1 INTRODUCTION

#### 1.1 STUDY DESIGN

This study is a multi-center, 24-week treatment, parallel group, double-blind, randomized, placebo-controlled study to evaluate the use of dupilumab in participants with prurigo nodularis (PN) inadequately controlled on topical prescription therapies or when those therapies are not advisable. The study will assess the effect of dupilumab on itch improvement as well as its effect on PN lesions, on participants' health-related quality of life (HRQoL), anxiety and depression, sleep quality, skin pain, and overall health status.

After 2-4 weeks of screening, participants will be centrally randomized using a permuted block randomization schedule via Interactive Voice Response System/Interactive Web Response System (IVRS/IWRS) in a 1:1 randomization ratio to dupilumab 300 mg q2w or matching placebo. Randomization will be stratified by documented history of atopy (atopic or non-atopic), stable use of topical corticosteroids (TCS)/ topical calcineurin inhibitors (TCI) (yes or no), and country/territory code.

A total of approximately 150 participants will be randomized to two treatment arms (75 participants/arm). The number of participants with active mild AD upon study entry will represent up to 10% of the atopic participants. Both the atopic and the non-atopic PN populations will each be capped at 60% of the total enrolled population.

The study duration consists of the following periods:

- Screening period (2-4 weeks)
- Randomized IMP intervention period (24 weeks)
- Follow-up period (12 weeks)

#### 1.2 OBJECTIVE AND ENDPOINTS

Table 2 - Objectives and endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| <ul> <li>To demonstrate the efficacy of dupilumab on itch<br/>response in participants with PN, inadequately<br/>controlled on topical prescription therapies or<br/>when those therapies are not advisable.</li> </ul> | <ul> <li>Proportion of participants with improvement<br/>(reduction) in worst-itch numeric rating scale (WI-NRS)<br/>by ≥4 from baseline to Week 12.</li> </ul> |
| Secondary | |
| <ul> <li>To demonstrate the efficacy of dupilumab on<br/>additional itch endpoints in participants with PN,<br/>inadequately controlled on topical prescription</li> </ul> | <ul> <li>Proportion of participants with improvement<br/>(reduction) in WI-NRS by ≥4 from baseline to Week 24<br/>[Key secondary endpoint].</li> </ul> |
| therapies or when those therapies are not advisable. | <ul> <li>Time to onset of effect on pruritus as measured by<br/>proportion of participants with an improvement<br/>(reduction) in WI-NRS by ≥4 from baseline during the<br/>24-week treatment period.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Change from baseline in WI-NRS at Week 24.</li> </ul> |
| | <ul> <li>Change from baseline in WI-NRS at Week 12.</li> </ul> |
| | <ul> <li>Percent change from baseline in WI-NRS at Week 24</li> </ul> |
| | Percent change from baseline in WI-NRS at Week 12 |
| | Percent change from baseline in WI-NRS at Week 4. |
| | Percent change from baseline in WI-NRS at Week 2. |
| | <ul> <li>Percent change from baseline in WI-NRS over time<br/>until Week 24.</li> </ul> |
| | <ul> <li>Proportion of participants with WI-NRS reduction ≥4 a<br/>Week 4.</li> </ul> |
| | <ul> <li>Proportion of participants with WI-NRS reduction</li> </ul> |
| | ≥4 over time until Week 24 <sup>a</sup> . |
| | <ul> <li>Onset of action in change from baseline in WI-NRS<br/>(first p &lt;0.05 difference from placebo in the daily<br/>WI-NRS that remains significant at subsequent</li> </ul> |
| | measurements) until Week 12 <sup>b</sup> . |
| <ul> <li>To demonstrate efficacy of dupilumab on skin<br/>lesions of PN.</li> </ul> | <ul> <li>Proportion of participants with Investigator's Global<br/>Assessment 0 or 1 score for PN-Stage (IGA PN-S) at<br/>Week 24 [Key secondary endpoint].</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-S 0 or 1 score<br/>at Week 12.</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-S 0 or 1 score<br/>at Week 8<sup>c</sup>.</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-S 0 or 1 score<br/>at Week 4<sup>c</sup>.</li> </ul> |
| | Change from baseline in IGA PN-S score at Week 24 |
| | Change from baseline in IGA PN-S score at Week 12 |
| | Change from baseline in IGA PN-S score at Week 8. |
| | Change from baseline in IGA PN-S score at Week 4. |
| | <ul> <li>Proportion of participants with Investigator's Global<br/>Assessment 0 or 1 score for PN-Activity (IGA PN-A) a<br/>Week 24.</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-A 0 or 1 score<br/>at Week 12.</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-A 0 or 1 score<br/>at Week 8.</li> </ul> |
| | <ul> <li>Proportion of participants with IGA PN-A 0 or 1 score<br/>at Week 4.</li> </ul> |
| <ul> <li>To demonstrate efficacy of dupilumab on both<br/>itch as well as skin lesions within the same<br/>participant</li> </ul> | <ul> <li>Proportion of participants with both an improvement<br/>(reduction) in WI-NRS by ≥4 from baseline to Week 2<br/>and an IGA PN-S 0 or 1 score at Week 24 (key<br/>secondary endpoint for US and US reference<br/>countries only)</li> </ul> |
| To demonstrate the improvement in health-<br>related quality of life (HRQoL). | Change from baseline in HRQoL, as measured by<br>Dermatology Life Quality Index (DLQI) to Week 24. |

| | Objectives | Endpoints |
|---|---|---|
| | | <ul> <li>Change from baseline in HRQoL, as measured by<br/>DLQI to Week 12.</li> </ul> |
| • | To evaluate safety outcome measures. | <ul> <li>Percentage of participants experiencing treatment-<br/>emergent adverse events (TEAEs) or serious adverse<br/>events (SAEs) from baseline through Week 24.</li> </ul> |
| • | To evaluate immunogenicity of dupilumab. | <ul> <li>Incidence of treatment-emergent antidrug antibodies<br/>(ADA) against dupilumab over time.</li> </ul> |
| Tertia | ry/exploratory | |
| • | To demonstrate a reduction in the use of rescue medication and systemic immunosuppressant | Use of high potency or superpotent TCS rescue<br>medication through Week 24 |
| | | <ul> <li>Use of systemic immunosuppressants through<br/>Week 24, constituting treatment failure</li> </ul> |
| • | To evaluate exploratory outcome measures | <ul> <li>Change from baseline in Hospital Anxiety and<br/>Depression Scale (HADS) total score to Week 24.</li> </ul> |
| | | <ul> <li>Change from baseline in EQ5D-5L to Week 24.</li> </ul> |
| | | <ul> <li>Change from baseline in skin Pain numeric rating<br/>scale (NRS) to Week 4, Week 8, Week 12, and<br/>Week 24, respectively.</li> </ul> |
| | | <ul> <li>Change from baseline in Sleep NRS to Week 4,<br/>Week 8, Week 12, and Week 24, respectively.</li> </ul> |
| | | <ul> <li>Missed school/work days through Week 24.</li> </ul> |
| | | <ul> <li>Incidence of skin-infection TEAEs (excluding herpetic<br/>infections) through Week 24.</li> </ul> |
| • | To evaluate the efficacy of dupilumab on skin lesions using a modified PAS 5-item questionnaire | <ul> <li>Proportion of participants who achieve ≥75% healed<br/>lesions from Prurigo Activity Score (PAS) at Week 4,<br/>Week 8, Week 12, and Week 24, respectively.</li> </ul> |
| | | <ul> <li>Change from baseline in exact number of lesions in<br/>representative area (as determined from PAS) at<br/>Week 4, Week 8, Week 12, and Week 24,<br/>respectively.</li> </ul> |
| • | To evaluate the efficacy of dupilumab on other PN endpoints | <ul> <li>Change from baseline in Participant Global Impression<br/>of Severity (PGIS) of PN to Week 4, Week 8,<br/>Week 12, and Week 24, respectively.</li> </ul> |
| | | <ul> <li>Participant Global Impression of Change (PGIC) of P<br/>at Week 4, Week 8, Week 12, and Week 24,<br/>respectively.</li> </ul> |
| PK | | |
| • | To evaluate pharmacokinetic (PK) and pharmacodynamic (PD) outcome measures | <ul> <li>Serum functional dupilumab concentrations and PK profile.</li> </ul> |
| | | Pharmacodynamic response for selected biomarkers (total IgE). White Will NRS reduction 24 between during and placebo will be |

a The early onset for significant change in the proportion of responders with WI-NRS reduction ≥4 between dupilumab and placebo will be claimed at Week xx if the p-value for Week xx is <0.05 and the remaining timepoints also have nominal p-value ≤0.05 until Week 12.

b The early onset for significant change in WI-NRS from baseline between dupilumab and placebo will be claimed at Week xx if the p-value for Week xx is <0.05 and the remaining timepoints also have nominal p-value ≤0.05 until Week 12.

c The early onset for reaching IGA PN-S(0,1) between dupilumab and placebo will be claimed at Week xx if the p-value for Week xx is <0.05 and the remaining timepoints also have nominal p-value ≤0.05 until Week 12.

## 1.2.1 Estimands

The primary estimands defined for main endpoints are summarized in below Table 3. More details are provided in Section 4.

Table 3 - Summary of primary estimand for main endpoints

| | Estimands | | | |
|---|---|---|---|---|
| Endpoint Category | Endpoint(s) <sup>a</sup> | Population | Intercurrent event(s) strategy and missing data handling | Population-level summary |
| Primary objective: To der therapies are not advisab | | oilumab on itch re | sponse in participants with PN, inadequately controlled on topical prescription ther | rapies or when those |
| Primary endpoint | Proportion of participants | ITT | The intercurrent events will be handled as follows: | CMH test adjusted by |
| | with improvement<br>(reduction) in worst-itch | | Discontinuation of study treatment before Week 12: Off-study treatment data up | documented history of atopy (atopic or non- |
| | numeric rating scale | | to Week 12 will be included in the analysis (treatment policy strategy). | atopic), stable use of |
| | (WI-NRS) by ≥4 from<br>baseline to Week 12 | | Taking the prohibited medications/procedures and/or rescue medications <sup>b</sup> prior | TCS/TCI (yes or no), region (countries |
| | | | to Week 12: Participants will be considered as non-responders (composite | combined), and |
| | | | strategy). | baseline antidepressant use (yes or no). |
| | | | In addition, the missing data imputation rules are as follows: | 200 (j 00 cio). |
| | | | <ul> <li>Having missing data at Week 12: Participants will be considered as non-<br/>responders.</li> </ul> | |

| | | | Estimands | |
|---|---|---|---|---|
| Endpoint Category | Endpoint(s) <sup>a</sup> | Population | Intercurrent event(s) strategy and missing data handling | Population-level summary |
| Secondary objective: To owner those therapies are | | dupilumab on add | itional itch endpoints in participants with PN, inadequately controlled on topical pr | escription therapies or |
| Secondary endpoint | Time to onset of effect on pruritus as measured by proportion of participants with an improvement (reduction) in WI-NRS by ≥4 from baseline during the 24-week treatment period | ITT | <ul> <li>Discontinuation of study treatment before Week 24: Off-study treatment data up to Week 24 will be included in the analysis (treatment policy strategy).</li> <li>Taking the prohibited medications/procedures and/or rescue medications<sup>b</sup> prior to Week 24: Analyses will be censored at Week 24 (composite strategy).</li> <li>In addition, the missing data imputation rules are as follows:</li> <li>Discontinuing the study follow-up before Week 24: Analyses will be censored at the time of last WI-NRS assessment.</li> </ul> | This time-to-event endpoint will be analyzed using the Cox proportional hazards model, including intervention group, documented history of atopy (atopic or nonatopic), stable use of TCS/TCI (yes or no), region (countries combined), and baseline antidepressant use (yes or no). The hazards ratio, its 95% confidence interval and p-value will be reported. Kaplan-Meier curves will be also provided. |

| | | | Estimands | |
|---|---|---|---|---|
| Endpoint Category | Endpoint(s) <sup>a</sup> | Population | Intercurrent event(s) strategy and missing data handling | Population-level summary |
| Secondary endpoint | Change from baseline in WI-NRS at Week 24 | ITT | <ul> <li>The intercurrent events will be handled as follows:</li> <li>Discontinuing the study treatment: all data collected following schedule after treatment discontinuation will be used in the analysis (treatment policy strategy).</li> <li>Taking the prohibited medications/procedures and/or rescue medications<sup>b</sup> prior to Week 24: data will be set to missing values after the medication usage, and the participant's worst postbaseline value on or before the time of the medication usage will be used to impute missing endpoint value (for participants whose postbaseline values are all missing, the participant's baseline will be used to impute the missing endpoint value) (hypothetical strategy)</li> <li>In addition, the missing data imputation rules are as follows:</li> <li>After discontinuation of the study treatment due to lack of efficacy prior to Week 24: WOCF approach will be used to impute missing data if needed<sup>2</sup>.</li> <li>After discontinuation of the study treatment due to reasons other than lack of efficacy prior to Week 24: multiple imputation (MI) approach will be used to impute missing endpoint value, and this multiple imputation will use all participants excluding participants who have taken the prohibited medications and/or rescue medications prior to Week 24 and excluding participants who discontinue due to lack of efficacy prior to Week 24.</li> </ul> | ANCOVA model with intervention group, documented history of atopy (atopic or nonatopic), stable use of TCS/TCI (yes or no), region (countries combined), baseline antidepressant use (yes or no), and relevant baseline measurement as covariates is used. Statistical inference obtained from all imputed data by ANCOVA model will be combined using Rubin's rule. |

a Additional secondary objectives/endpoints are not included in this table but would be handled with a similar strategy as the endpoint type (ie continuous, proportion, time-to-event) at other weeks

b Prohibited medications and/or rescue medications are listed in Table 5.

## 2 SAMPLE SIZE DETERMINATION

The primary endpoint is the proportion of participants with WI-NRS reduction of ≥4 from baseline to Week 12. By assuming the response rate is in the placebo and dupilumab arms, respectively, 56 participants/arm will provide 90% power to detect the difference of between dupilumab and placebo with Fisher exact test at 2-sided level of 0.05. Assuming 15% drop out during the 12 weeks of treatment, the target is to randomize 75 participants/arm with a cap of up to 10% of participants in the atopic population having active mild AD.

The assumptions were based on the effect of dupilumab versus placebo in WI-NRS reduction ≥4 at Week 16 observed in participants with moderate to severe AD as seen in studies of AD-1334 (Solo1) and AD-1416 (Solo2).

Approximately 150 participants will be randomized to dupilumab or placebo in a 1:1 ratio with stratification factors of documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), and country/territory code. Both the atopic and the non-atopic PN population will be capped at 60% of the total enrolled population.

The sample size calculation was performed using SAS 9.4 power procedure.

# 3 ANALYSIS POPULATIONS

The following populations for analyses are defined:

Table 4 - Populations for analyses

| Population | Description |
|---|---|
| Screened | All participants who sign the ICF. |
| Randomized | The randomized population includes all participants with a treatment kit number allocated and recorded in the interactive response technology (IRT) database, and regardless of whether the treatment kit was used or not. |
| | Participants treated without being randomized will not be considered randomized and will not be included in any efficacy population. |
| Intent-to-treat (ITT) | All randomized participants analyzed according to the intervention group allocated by randomization regardless if treatment kit is used or not |
| Efficacy | The ITT population |
| Safety | All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants will be analyzed according to the intervention they actually received. |
| | Randomized participants for whom it is unclear whether they took the study medication will be included in the safety population as randomized. |
| | For participants who accidentally receive different treatment from the planned, the actual intervention allocation for as-treated analysis will be the dupilumab group. |
| | The PD analyses will be performed on the safety population. |
| Pharmacokinetic (PK) | The PK population includes all participants in the safety population with at least one non-<br>missing result for functional dupilumab concentration in serum after first dose of the study<br>treatment. Participants will be analyzed according to the intervention actually received. |
| Antidrug antibody (ADA) | ADA population includes all participants in the safety population who have at least one non-missing ADA result after first dose of the study treatment. Participants will be analyzed according to the intervention actually received. |

ADA: antidrug antibody; ICF: informed consent form; ITT: intent to treat; PD: pharmacodynamics: PK: pharmacokinetic.

Participants exposed to study intervention before or without being randomized will not be considered randomized and will not be included in any analysis population. The safety experience of these participants will be reported separately.

Randomized participants for whom it is unclear whether they took the study intervention will be considered as exposed and will be included in the safety population as randomized.

For any participant randomized more than once, only the data associated with the first randomization will be used in any analysis population. The safety experience associated with any later randomization will be reported separately.

For participants receiving more than one study intervention (placebo and dupilumab) during the study, the intervention group for as-treated analysis will be the dupilumab group.

Statistical Analysis Plan SAR231893 (REGN668) - EFC16460 - dupilumab 08-Aug-2021 Version number: 2

Regarding the COVID-19 pandemic, additional summaries by COVID-19 subgroups (i.e., impacted by the COVID-19 pandemic and NOT impacted by the COVID-19 pandemic) will be provided to assess the impact of COVID-19 on treatment effect. Participants impacted by the COVID-19 pandemic are defined as randomized participants with any critical or major deviation related to COVID-19 or who permanently discontinued study intervention or study due to COVID-19.

## 4 STATISTICAL ANALYSES

#### 4.1 GENERAL CONSIDERATIONS

In general, continuous data will be summarized using the number of observations available, mean, standard deviation (SD), median, minimum, and maximum. Categorical and ordinal data will be summarized using the count and percentage of participants.

The baseline value of efficacy parameters is defined as the last available value before randomization and prior to the first dose of study medication unless below eDiary data (WI-NRS, skin Pain-NRS and Sleep-NRS) score or otherwise specified.

The baseline for weekly average WI-NRS (skin Pain-NRS and Sleep-NRS) score is defined as the average of daily non-missing scores obtained during the 7 days prior to randomization.

The baseline value of the other parameters is defined as the last available value prior to the first dose of investigational medicinal product (IMP) if the participant is treated, or the last available value up to randomization if the participant is not exposed to IMP.

## Observation period

The observation period will be divided into 4 segments:

- The **pre-treatment period** is defined as the period up to first IMP administration.
- The **treatment-emergent (TE) period** is defined as the period from the first IMP administration to the last IMP administration + 98 days. The treatment-emergent period includes the following 2 periods:
  - The **on-treatment period** is defined as the period from the first IMP administration to the last administration of the IMP + 14 days
  - The **residual treatment period** is defined as the period from the end of the ontreatment period to the end of the treatment-emergent period.
- The **post-treatment period** is defined as the period from the end of the treatmentemergent period.

The on-study observation period is defined as the time from start of intervention until the end of the study defined as the status date collected on e-CRF page "Completion of End of Study".

#### 4.2 PARTICIPANT DISPOSITIONS

The number (%) of participants included in each of the analysis populations listed in Table 4 will be summarized.

Screen failures are defined as participants who consent to participate in the study but are not subsequently randomized. The number (%) of screen failures and reasons for screen failures will be provided in the screened population.

The number (%) of participants in the following categories will be provided:

- Randomized participants
- Randomized but not exposed participants
- Randomized and exposed participants
- Participants who completed the study treatment period as per protocol
- Participants who did not complete the study treatment period as per protocol and discontinued study treatment prior to Week 12 by main reason for permanent intervention discontinuation including due to COVID-19
- Participants who did not complete the study treatment period as per protocol and discontinued study treatment prior to Week 24 by main reason for permanent intervention discontinuation including due to COVID-19
- Participants who completed the study period as per protocol
- Participants who did not complete the study period as per protocol and discontinued study by main reason for study discontinuation including due to COVID-19.
- Vital status at last study contact

The number (%) of exposed and not randomized participants will also be summarized.

In addition, the number (%) of participants screened, screened-failed, randomized, with permanent intervention discontinuation and with early study discontinuation will be provided by country and site.

#### Protocol deviations

Critical and major protocol deviations (automatic or manual) will be summarized in the randomized population and according to COVID-19 impact (i.e. deviations related to the COVID-19 pandemic). In addition, deviations potentially impacting the primary endpoint analysis will be summarized.

## 4.3 PRIMARY ENDPOINT(S) ANALYSIS

#### 4.3.1 Definition of endpoint(s)

The primary endpoint for this study is the proportion of participants with improvement (reduction) in worst-itch numeric rating scale (WI-NRS) by  $\geq 4$  from baseline to Week 12.

WI-NRS is a patient-reported outcome (PRO) comprised of a single item rated on a scale from 0 ("No itch") to 10 ("Worst imaginable itch"). Participants are asked to rate the intensity of their worst pruritus (itch) over the past 24 hours using this scale.

The weekly average WI-NRS score at each week, which is defined as the average of daily non-missing scores within the week window of each week (see Section 5.4), will be used for analyses.

For efficacy analysis, Table 5 presents the prohibited and rescue medications/procedures which will be considered as intercurrent events if the last column indicates as "Yes" and therefore be handled in the estimands for endpoints defined in Table 3.

Table 5 - Prohibited medications/procedures and rescue medications that impact efficacy

| Medication/procedure | Comment | Data to be set as non-<br>responder after taking<br>medication in the main<br>statistical analysis<br>(Yes/No) <sup>a</sup> / Selection<br>criteria |
|---|---|---|
| Prohibited medications/procedures | | |
| Systemic immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon gamma, Janus kinase inhibitors, azathioprine, methotrexate, hydroxychloroquine, dapsone, sulfasalazine, colchine, etc) | IMP to be discontinued | Yes (CDG <sup>b</sup> Immunosuppressant drugs Narrow and SDG <sup>b</sup> Corticosteroids Narrow) |
| Other monoclonal antibodies (that are biological response modifiers). | IMP to be discontinued | Yes (SDG <sup>b</sup> Monoclonal antibodies Narrow) |
| Phototherapy, including tanning beds. | IMP to be discontinued | Yes (CMQ <sup>b</sup> HLT Phototherapies, CMQ <sup>b</sup> Tanning_single PT) |
| Naltrexone or other opioid antagonist | IMP to be discontinued | Yes (SDG <sup>b</sup> Analgesia producing opioids NARROW) |
| Gabapentin, pregabalin, and thalidomide | IMP to be discontinued | Yes (CDG <sup>b</sup> Gabapentin mono and multi ingredients, Pregabalin mono and multi ingredients, or Thalidomide mono and multi ingredients) |
| Paroxetine, fluvoxamine or other SSRIs. | No IMP discontinuation, see requirement in the footnote | Yes <sup>c,d</sup> (CDG <sup>b</sup> N06AB selective serotonin reuptake inhibitors) |
| SNRIs. | No IMP discontinuation, see requirement in the footnote | Yes <sup>c,d</sup> (CDG <sup>b</sup> serotonin and norepinephrine reuptake inhibitors) |
| Amitriptyline or other tricyclic or tetracyclic antidepressants | No IMP discontinuation, see requirement in the footnote | Yes <sup>c,d</sup> (CDG <sup>b</sup> N06AA non-selective monoamine reuptake inhibitors) |
| Intralesional corticosteroid injections and cryotherapy. | No IMP discontinuation | Yes <sup>d</sup> (CMQ <sup>b</sup> Injection_single pt,<br>cryotherapy or skin cryotherapy<br>PT) |
| Sedating antihistamine | No IMP discontinuation | Yes <sup>d,e</sup> (CDG <sup>b</sup> sedating antihistamines) |
| Non-sedating antihistamine if used specifically for the treatment of itch secondary to AD or PN | No IMP discontinuation | Yes <sup>d.e</sup> (CDG <sup>b</sup> non-sedating antihistamines) |

| Medication/procedure | Comment | Data to be set as non-<br>responder after taking<br>medication in the main<br>statistical analysis<br>(Yes/No) <sup>a</sup> / Selection<br>criteria |
|---|---|---|
| Rescue medications | | |
| Dermatological preparations of high potency or superpotent TCS and TCI | No IMP discontinuation | Yes <sup>d</sup> (CDG <sup>b</sup> calcineurin inhibitors and corticosteroids narrow, Ticked 'RESCUE THERAPY' in CRF page) |

- a. When yes, the estimand for the intercurrent event handling strategy will be as follows: hypothetical for continuous endpoints, and composite for responder and time-to-event endpoints. When no, a treatment policy strategy will be applied.
- b. CDG=company drug groupings, CMQ=company MedDRA query, SDG= Standardized drug groupings.
- c. Only if the antidepressant is initiated during the study or its dose is increased from baseline provided that medication was taken at least 3 months prior to screening.
- d. As per medical adjudication, see Appendix 7 for details.
- e. Only if the medication is initiated at Week 12 or Week 24, or the dose is increased from Week 11 to Week 12 or from Week 23 to Week 24.

Blinded review of prohibited/rescue treatment (medication or procedure) based on Table 5 and a pre-specified algorithm (Appendix 7) will be implemented before database locks by considering the type of medication or procedure, indication, timing, frequency and the potential impact of the use of the prohibited medications/procedures and rescue medications.

## 4.3.2 Main analytical approach

The primary estimand for the primary endpoint is the treatment policy/composite approach as defined in Table 3.

The primary analysis population for the efficacy endpoints will be the ITT population.

The following null hypothesis H0 and alternative hypothesis H1 will be tested for dupilumab against placebo:

- H0: No treatment difference between dupilumab and placebo.
- H1: There is a treatment difference between dupilumab and placebo

The primary analysis will be conducted by using Cochran–Mantel–Haenszel test (CMH) test adjusted by documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region, and baseline anti-depressant use (yes or no). Comparisons of the response rates between dupilumab and placebo will be derived. In addition, odds ratio and response rate difference as well as the corresponding 95% confidence intervals (CI) will be provided along with the p-values.

As defined in Table 3 for participants discontinuing the study treatment before Week 12, their off-study treatment values measured up to Week 12 will be included in the analysis. Participants taking the prohibited medications/procedures and/or rescue medications (see Table 5) prior to Week 12 or having missing data at Week 12 will be considered non-responders.

#### 4.3.3 Sensitivity analysis

For the primary estimand for the primary endpoint, no sensitivity analysis will be performed. However, three supplementary analyses will be performed as described in the section below.

#### 4.3.4 Supplementary analyses

The following supplementary analyses will be performed:

As-observed analysis (including all data after taking the prohibited and/or rescue medications)

The data collected after taking all prohibited medications and/or rescue medications will be included in the supplementary analysis to evaluate the robustness of the primary analysis results with respect to the method of handling data while taking the prohibited medications (e.g. treatment policy strategy). In addition, for participants discontinuing the study treatment before Week 12, their off-study treatment values measured up to Week 12 will be included in the analysis. The participants having missing data at Week 12 regardless of reason(s) will be considered non-responders at that timepoint.

Hybrid method analysis (the worst-observation carried forward (WOCF) and multiple imputation (MI))

In the primary analysis of change from baseline in WI-NRS (continuous variable) at Week 12, the hybrid method of the WOCF and MI will be used (see Section 4.4.2). Similar to the continuous variable, the same imputation method will be used in the analysis of the proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 12, which is consistent for the intercurrent event strategy and missing data handling in the binary variables and continuous variable. That is, after the imputation of continuous WI-NRS data at Week 12 using the hybrid method of the WOCF and MI (see Section 4.4.2), responders will be defined as participants with improvement in WI-NRS by ≥4 from baseline to Week 12 in each of the imputed datasets with about 40 imputations, and then the CMH test adjusted by documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region, and baseline antidepressant use (yes or no) will be used. Statistical inference obtained from all imputed data will be combined using Rubin's rule.

#### Tipping point analysis

The intercurrent events will be handled as follows:

- Discontinuation of study treatment before Week 12: Off-study treatment data up to Week 12 will be included in the analysis (treatment policy strategy).
- Taking the prohibited medications/procedures and/or rescue medications prior to Week 12: Data after the intercurrent events will be censored and then imputed with the below tipping point method

In addition, the missing data imputation rules are as follows:

 Having missing data at Week 12: Data will be imputed with the following tipping point method.

## Tipping point method:

- A sequence of analyses will be performed with the adjustment to artificially decrease the response rate in the dupilumab group and increase the response rate in the placebo group with a fixed and definite set of values for data imputation.
- For each combination of increasing response rate in placebo and decreasing response rate in dupilumab, multiple imputed datasets will be generated and analyzed using CMH test. The results obtained from multiple imputed datasets will be combined to generate statistical inference, i.e. p-value and treatment difference between 2 treatment groups.
- A "tipping point" will be identified while the result is no longer statistically significant (i.e. p-value >0.05).

## 4.3.5 Subgroup analyses

To assess the homogeneity of the treatment effect across various subgroups, analyses will be performed on the primary endpoint across the following subgroups (categories with fewer than 5 participants may be combined with other categories):

- Age group ( $<65, \ge 65$  years)
- Gender (Male, Female)
- Region
- Territory
- Race (Caucasian/White, Black/of African descent, Asian/Oriental, Others)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Baseline weight ( $<60, \ge 60 < 90, \ge 90 \text{ kg}$ )
- Baseline BMI ( $<25, \ge 25 <30, \ge 30 \text{ kg/m}^2$ )
- Participants without a current diagnosis of AD
- History of atopy (atopic or non-atopic)
- Stable use of TCS/TCI (yes or no)
- Antidepressant use (yes or no) at baseline
- Baseline IGA PN-S moderate versus severe (3 vs. 4)
- Participants who have not been impacted by COVID-19 vs impacted by COVID-19 (for
  participants who have been impacted by the COVID-19, the efficacy data will be
  descriptive only if the number of participants is not enough to perform statistical tests.
  Participants impacted by the COVID-19 pandemic are defined as randomized participants
  with any critical or major deviation related to COVID-19 or who permanently
  discontinued study intervention or study due to COVID-19.)

To test the interaction between intervention and subgroup factor, a logistic regression model incorporating subgroup-by-treatment interaction will be built for each subgroup factor except the subgroup of participants without a current diagnosis of AD (very few AD participants will be excluded). The model will include all the covariates in the main statistical model plus the subgroup variable and the subgroup-by-treatment interaction. A p-value for the test of interaction will be provided.

In each subgroup, the treatment effects for the primary endpoint will be provided, as well as the corresponding 95% CI, using the same method as applied to the primary analysis. Forest plots will be provided.

## 4.4 SECONDARY ENDPOINT(S) ANALYSIS

The weekly average skin Pain-NRS or Sleep-NRS score at each week, which is defined as the average of non-missing daily scores within the week window of each week (see Section 5.4), will be used for analyses.

## 4.4.1 Key/Confirmatory secondary endpoint(s)

#### 4.4.1.1 Definition of endpoint(s)

The key secondary endpoints are:

- Proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24, and
- Proportion of participants with IGA PN-S 0 or 1 score at Week 24.

In addition, for US and US reference countries only, there is another key secondary endpoint:

• Proportion of participants with both an improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24 and an IGA PN-S 0 or 1 score at Week 24.

## Investigator's global assessment for prurigo nodularis (IGA PN)

The IGA PN is a clinician-reported outcome (ClinRO) that allows clinicians to assess the activity of PN (IGA PN-A) using a 5-point scale from 0 (clear) to 4 (severe); and the stage of the disease (IGA PN-S) using a 5-point scale from 0 (clear) to 4 (severe).

#### 4.4.1.2 Main analytical approach

For the key secondary efficacy endpoints, the analysis will be conducted by using CMH test adjusted by documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region, and baseline anti-depressant use (yes or no). The same estimand, i.e., intercurrent event strategy and missing data handling method, as the primary endpoint, by replacing Week 12 with Week 24, is used.

The same supplementary and subgroup analyses used for the primary endpoint will also be performed for the key secondary efficacy endpoints.

## 4.4.2 Supportive secondary endpoint(s)

The other secondary endpoints are as follows:

- Proportion of participants with WI-NRS reduction ≥4 over time until Week 24.
- Proportion of participants with WI-NRS reduction ≥4 at Week 4
- Proportion of participants with IGA PN-S 0 or 1 score at Week 12
- Proportion of participants with IGA PN-S 0 or 1 score at Week 8
- Proportion of participants with IGA PN-S 0 or 1 score at Week 4
- Proportion of participants with IGA PN-A 0 or 1 score at Week 24
- Proportion of participants with IGA PN-A 0 or 1 score at Week 12
- Proportion of participants with IGA PN-A 0 or 1 score at Week 8
- Proportion of participants with IGA PN-A 0 or 1 score at Week 4
- Time to onset of effect on pruritus as measured by proportion of participants with an improvement (reduction) in WI-NRS by ≥4 from baseline during the 24-week treatment period
- Change from baseline in WI-NRS at Week 24
- Change from baseline in WI-NRS at Week 12
- Percent change from baseline in WI-NRS at Week 24
- Percent change from baseline in WI-NRS at Week 12
- Percent change from baseline in WI-NRS at Week 4
- Percent change from baseline in WI-NRS at Week 2
- Percent change from baseline in WI-NRS over time until Week 24.
- Onset of action in change from baseline in WI-NRS (first p <0.05 difference from placebo in the daily WI-NRS that remains significant at subsequent measurements) until Week 12
- Change from baseline in IGA PN-S score at Week 24
- Change from baseline in IGA PN-S score at Week 12
- Change from baseline in IGA PN-S score at Week 8
- Change from baseline in IGA PN-S score at Week 4
- Change from baseline in HRQoL, as measured by Dermatology Life Quality Index (DLQI) to Week 24

 Change from baseline in HRQoL, as measured by Dermatology Life Quality Index (DLQI) to Week 12

## Dermatology life quality index (DLQI)

The DLQI is a PRO developed to measure dermatology-specific HRQoL in adult participants. The instrument comprises 10 items assessing the impact of skin disease on participants' HRQoL over the previous week. The items cover symptoms, leisure activities, work/school or holiday time, personal relationships including intimate, the side effects of treatment, and emotional reactions to having a skin disease. It is a validated questionnaire used in clinical practice and clinical trials. Response scale is a 4-point Likert scale (0 = "not at all" and 3 = "very much") for nine items. The remaining one item about work/studying asks whether work/study has been prevented and then (if "No") to what degree the skin condition has been a problem at work/study; the item is rated on a 3-point Likert scale ("Not at all" to "A lot"). Overall scoring ranges from 0 to 30, with a high score indicative of a poor HRQoL.

#### Time-to-event secondary efficacy endpoint

Time to first onset of effect on pruritus defined as an improvement (reduction) in WI-NRS by ≥4 from baseline during the 24-week treatment period will be analyzed using the Cox proportional hazards model, including treatment, documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region, and baseline anti-depressant use (yes or no). The hazards ratio, its 95% confidence interval and p-value will be reported. Kaplan-Meier curves will be also provided.

For time to first WI-NRS response (WI-NRS by  $\geq 4$  from baseline), participants who receive the prohibited medications and/or rescue medications (see Table 5), data prior to start of the medications will be used, but after medication start, the participants' data will not be used and they will be censored at Week 24 (i.e. Day 172). For other participants, all available data up to Week 24 (i.e. Day 172) including those collected during the off-treatment period will be used. Participants without events will be censored at Day 172 or their last WI-NRS assessment date if discontinued from the study, whichever is earlier.

#### Secondary efficacy endpoints that measure binary responses

Secondary efficacy endpoints that measure binary responses will be analyzed in the same fashion as the primary endpoint using primary statistical model.

#### Continuous secondary efficacy endpoints

The primary estimand for continuous secondary efficacy endpoints is defined in Table 3 and will be analyzed using an analysis of covariance (ANCOVA) model with intervention group, documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region (countries combined), baseline antidepressant use (yes or no), and relevant baseline measurement as covariate, with intercurrent event strategy and missing data handling as defined as in Table 3. Specifically, data of participants taking the prohibited medications/procedures and/or rescue medications will be set to missing after the medication usage, and the worst postbaseline value on

or before the time of the medication usage will be used to impute missing endpoint value (for participants whose postbaseline values are all missing, the baseline will be used to impute). Participants who discontinue the treatment prematurely are encouraged to follow the planned clinical visits and in those participants who did not take the prohibited medications/procedures and/or rescue medications, all data collected after treatment discontinuation will be used in the analysis. For these participants, missing data may still happen despite all efforts have been tried to collect the data after treatment discontinuation. For participants who discontinue due to lack of efficacy, all data collected after discontinuation will be used in the analysis, and a WOCF approach will be used to impute missing data if needed. For participants who discontinued not due to lack of efficacy, a multiple imputation (MI) approach will be used to impute missing endpoint value, and this MI method will use all participants excluding participants who have taken the prohibited medications/procedures and/or rescue medications prior to timepoint of endpoint of interest and excluding participants who discontinue due to lack of efficacy.

Each of the imputed complete data will be analyzed by fitting an ANCOVA model as described above. The imputation number will be about 40. Statistical inference obtained from all imputed data will be combined using Rubin's rule. Descriptive statistics including number of participants, mean, standard error, and least squares (LS) mean changes (and standard error) will be provided. In addition, difference of the dupilumab group against placebo in LS means and the corresponding 95% confidence intervals (CI) will be provided along with the p-values.

See Section 5.5 for the sample SAS code for the imputation and the analysis.

For the endpoint of percent change from baseline in WI-NRS at week 24, we will also perform an as-observed plus multiple imputation supplementary analysis as described below.

The data collected after taking all prohibited medications and/or rescue medications will be included in the supplementary analysis to evaluate the robustness of the primary analysis results with respect to the method of handling data while taking the prohibited medications (e.g. treatment policy strategy). In addition, for participants discontinuing the study treatment before Week 24, their off-study treatment values measured up to Week 24 will be included in the analysis. For participants having missing data at Week 24 regardless of reason(s), a multiple imputation (MI) approach will be used to impute the missing endpoint value.

#### 4.5 TERTIARY/EXPLORATORY ENDPOINT(S) ANALYSIS

## 4.5.1 Definition of endpoint(s)

The exploratory endpoints are as follows:

- Use of high potency or superpotent TCS rescue medication through Week 24
- Use of systemic immunosuppressant through Week 24, constituting treatment failure
- Change from baseline in Hospital Anxiety and Depression Scale (HADS) total score to Week 24
- Change from baseline in EQ-5D-5L Single Index score to Week 24

- Change from baseline in EQ-5D visual analog scale (VAS) to Week 24
- Change from baseline in skin Pain-NRS to Week 4, Week 8, Week 12, and Week 24, respectively
- Change from baseline in Sleep-NRS to Week 4, Week 8, Week 12, and Week 24, respectively
- Missed school/work days through Week 24
- Incidence of skin-infection TEAEs (excluding herpetic infections) through Week 24
- Proportion of participants who achieve ≥75% healed lesions from PAS at Week 4, Week 8, Week 12, and Week 24, respectively
- Change from baseline in exact number of lesions in representative area (as determined from PAS) at Week 4, Week 8, Week 12, and Week 24, respectively
- Change from baseline in Participant Global Impression of Severity (PGIS) of PN to Week 4, Week 8, Week 12, and Week 24 respectively
- Proportion of participants with PGIS score of "none" at Week 4, Week 8, Week 12, and Week 24 respectively
- Proportion of participants with PGIS score of "none" or "mild" at Week 4, Week 8, Week 12, and Week 24 respectively
- Participant Global Impression of Change (PGIC) of PN at Week 4, Week 8, Week 12, and Week 24, respectively
- Proportion of participants with PGIC score of "very much better" at Week 4, Week 8, Week 12, and Week 24 respectively
- Proportion of participants with PGIC score of "very much better" or "moderately better" at Week 4, Week 8, Week 12, and Week 24 respectively

#### Hospital anxiety and depression scale (HADS)

The HADS is a PRO instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes to a participant's emotional state. The HADS consists of 14 items, 7 each for anxiety and depression symptoms; possible scores range from 0 to 21 for each subscale. The following cut-off scores are recommended for both subscales:

- 0 to 7: normal
- 8 to 10: borderline abnormal (borderline case)
- 11 to 21: abnormal

## Euroqol 5 dimensions questionnaire (EQ-5D)

The Euroqol-5 dimensions (EQ-5D) is a standardized PRO measure of health status developed by the EuroQOL Group in order to provide a simple, generic measure of health for clinical and

economic appraisal. The EQ-5D consists of 2 parts: the descriptive system and the EQ visual analog scale (VAS). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of perceived problems: "no problem", "slight problems", "moderate problems", "severe problems" and "inability to do the activity". The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions; this results in a 1-digit number expressing the level for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labeled "best imaginable health state (100)" and "worst imaginable health state (0)". This information can be used as a quantitative measure of health outcome as judged by the individual respondents.

#### Skin Pain and sleep numeric rating scales (skin Pain-NRS, Sleep-NRS)

Participants will be asked to rate their worst skin pain in the past 24 hours using a 0 to 10 NRS, with 0 = No pain to 10 = Worst pain possible.

In addition, participants will be asked to rate their sleep quality on their past night upon awakening, using a 0 to 10 NRS, with 0 = Worst possible sleep and 10 = Best possible sleep.

Participants will complete the skin pain NRS and sleep quality NRS once a day.

## Prurigo activity score (PAS)

The PAS is a clinician-reported outcome (ClinRO) measurement. The original PAS questionnaire Version 0.9 consists of 7 items, developed by expert clinicians in PN.

A 5-item simplified version of the PAS will be used in the current study. Item 4 (exact number of pruriginous lesions in representative area) and Item 5b (percentage of healed prurigo lesions in all pruriginous lesions) will be used for analyses. In addition, Item 2 (number of prurigo lesions) may be used for analysis too.

# <u>Participant Global Impression of Change of disease (PGIC) and Participant Global Impression of Severity (PGIS)</u>

The PGIC is a one-item questionnaire that asks participants to provide the overall self-assessment of change in their PN overall on a 7-point scale, compared to just before participant started taking the study injection. Response choices are: 0 = "Very much better", 1 = "Moderately better", 2 = "A little better", 3 = "No change", 4 = "A little worse", 5 = "Moderately worse", 6 = "Very much worse".

The PGIS is a one-item questionnaire that asks participants to provide the overall self-assessment of their disease severity on a 4-point scale for the past week. Response choices are: 1 = "none", 2 = "Mild", 3 = "Moderate", 4 = "Severe".

## Missed school/work days

Participants who are employed or enrolled in school will be asked to report the number of sick leave/missed school days since the last study assessment.

## 4.5.2 Main analytical approach

Exploratory efficacy endpoints will be analyzed using the same methodology as secondary efficacy for similar data (continuous or proportion) except the endpoints below.

- Use of high potency or superpotent TCS rescue medication through Week 24
- Use of systemic immunosuppressant through Week 24, constituting treatment failure
- Missed school/work days through Week 24
- Incidence of skin-infection TEAEs (excluding herpetic infections) through Week 24

The number of participants and percentage with the events for these endpoints will be provided in observed cases. In addition, the time (week) to first event for those participants will also be analyzed using Kaplan-Meier method and the duration of the rescue medication use may be summarized if applicable.

An additional exploratory endpoint of time to first select prohibited/rescue medication that impact efficacy will be provided. This includes medications where WOCF will be applied (see Table 5).

#### 4.6 MULTIPLICITY ISSUES

The multiplicity procedure is proposed to control the overall type-I error rate for testing the primary and selected secondary endpoints. The overall alpha is 0.05. The comparisons with placebo will be tested based on the hierarchical order below at 2-sided  $\alpha = 0.05$ :

## **In US and US reference countries:**

- Proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 12.
- Proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24
- Proportion of participants with IGA PN-S 0 or 1 score at Week 24
- Proportion of participants with both an improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24 and an IGA PN-S 0 or 1 score at Week 24
- Proportion of participants with IGA PN-S 0 or 1 score at Week 12
- Percent change from baseline in WI-NRS at Week 24
- Change from baseline in HRQoL, as measured by Dermatology Life Quality Index (DLQI) to Week 24
- Change from baseline in skin Pain-NRS to Week 24

- Change from baseline in Sleep-NRS to Week 24
- Change from baseline in Hospital Anxiety and Depression Scale (HADS) total score to Week 24

# <u>In all other countries (including EU and EU reference countries, as well as China and Japan):</u>

- Proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 12.
- Proportion of participants with improvement (reduction) in WI-NRS by ≥4 from baseline to Week 24
- Proportion of participants with IGA PN-S 0 or 1 score at Week 24
- Percent change from baseline in WI-NRS at Week 24
- Proportion of participants with IGA PN-S 0 or 1 score at Week 12
- Change from baseline in HRQoL, as measured by Dermatology Life Quality Index (DLQI) to Week 24
- Change from baseline in skin Pain-NRS to Week 24
- Change from baseline in Sleep-NRS to Week 24
- Change from baseline in Hospital Anxiety and Depression Scale (HADS) total score to Week 24

The study is considered positive when the primary endpoint achieves statistical significance.

## 4.7 SAFETY ANALYSES

All safety analyses will be performed on the safety population as defined in Section 3, unless otherwise specified, using the following common rules:

- The analysis of the safety variables will be descriptive, and no testing is planned.
- Safety data in participants who do not belong to the safety population (e.g., exposed but not randomized) will be provided separately.

#### 4.7.1 Extent of exposure

The extent of IMP exposure will be assessed by the duration of IMP exposure and compliance and summarized within the safety population.

## **Duration of IMP exposure**

Duration of IMP exposure is defined as last dose date – first dose date + 14 days, regardless of unplanned intermittent discontinuations. Duration of IMP exposure will be summarized descriptively as a quantitative variable (number, mean, SD, median, minimum, and maximum). In addition, duration of treatment exposure will also be summarized categorically by numbers and percentages for each of the following categories and cumulatively according to these categories:

- >0 and <2 weeks
- >2 and <4 weeks
- >4 and <8 weeks
- >8 and <12 weeks
- >12 and <16 weeks
- >16 and ≤20 weeks
- >20 and ≤24 weeks
- >24 weeks and  $\leq 24$  weeks + 3 days
- > 24 weeks + 3 days

Additionally, the cumulative duration of treatment exposure will be provided, defined as the sum of the duration of treatment exposure for all participants, and will be expressed in participant years.

#### **Treatment compliance**

A given administration will be considered noncompliant if the participant did not take the planned dose as required by the protocol. No imputation will be made for participants with missing or incomplete data.

**Percentage of treatment compliance** for a participant will be defined as the number of administrations that the participant was compliant divided by the total number of administrations that the participant was planned to take from the first administration of IMP up to the actual last administration of IMP.

Treatment compliance will be summarized quantitatively and categorically: <80%,  $\ge80\%$ .

Cases of overdose (defined as at least twice the intended dose during an interval of less than 11 days) will be considered an AESI per dupilumab clinical programs and will be listed as such.

#### 4.7.2 Adverse events

#### General common rules for adverse events

All adverse events (AEs) will be coded to a lower-level term (LLT), preferred term (PT), high-level term (HLT), high-level group term (HLGT), and associated primary system organ class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA) version currently in effect at Sanofi at the time of database lock.

The AEs will be analyzed in the following 3 categories:

• Pre-treatment AEs: AEs that developed, worsened or became serious during the pre-treatment period.

- Treatment-emergent adverse events (TEAE)s: AEs that developed, worsened or became serious during the treatment-emergent period
- Post-treatment AEs: AEs that developed, worsened or became serious during the post-treatment period

Similarly, the deaths will be analyzed in the pre-treatment, treatment-emergent and post-treatment periods.

The primary focus of AE reporting will be on TEAEs. Pre-treatment and post-treatment AEs will be described separately.

An AE with incomplete or missing date/time of onset (occurrence, worsening, or becoming serious) will be classified as a TEAE unless there is definitive information to determine it is a pretreatment or a post-treatment AE.

If the assessment of the relationship to IMP is missing for an AE, this AE will be assumed as related to IMP. If the severity is missing for 1 of the treatment-emergent occurrences of an AE, the severity will be imputed with the maximal severity of the other occurrences. If the severity is missing for all the occurrences, the severity will be left as missing.

Multiple occurrences of the same event in the same participant will be counted only once in the tables within a treatment phase.

The AE tables will be sorted as indicated in Table 6.

Table 6 - Sorting of AE tables

| AE presentation | Sorting rules |
|---|---|
| SOC, HLGT, HLT and PT | By the internationally agreed SOC order and by alphabetic order of HLGTs, HLTs and PTs. |
| SOC, HLT and PT | By the internationally agreed SOC order and by alphabetic order of HLTs and PTs. |
| SOC and PT | By the internationally agreed SOC order and decreasing frequency of PTs <sup>a, b</sup> |
| SMQ/CMQ and PT | By decreasing frequency of SMQs/CMQs and PTs <sup>a</sup> |
| PT | By decreasing frequency of PTs <sup>a</sup> |

a Sorting will be based on the SAR231893 dupilumab group

#### Analysis of all adverse events

The overview of TEAE with the details below will be generated:

- Any TEAE
- Any severe TEAE
- Any treatment emergent SAE
- TEAE leading to death

b The table of all TEAEs presented by SOC and PT will define the presentation order for all other tables (eg, treatment-emergent SAE) presented by SOC and PT, unless otherwise specified.

- Any TEAE leading to permanent intervention discontinuation
- Any treatment emergent AESI
- Any treatment emergent other AE of interest grouping
- Any TEAE related to IMP

The AE summaries of Table 7 will be generated with number (%) of participants experiencing at least one event.

Table 7 - Analyses of adverse events

| Type of AE | MedDRA levels |
|---|---|
| All TEAE | Primary SOC, HLGT, HLT and PT |
| | Primary SOC and PT |
| | PT |
| | Primary and secondary SOC, HLGT, HLT and PT |
| Common TEAE (≥2% and 5% in any group) | Primary SOC and PT |
| TEAE related to IMP as per Investigator's judgment | Primary SOC, HLGT, HLT and PT |
| | Primary SOC and PT |
| TEAE by maximal intensity | Primary SOC and PT |
| Treatment emergent SAE | Primary SOC, HLGT, HLT and PT |
| | Primary SOC and PT |
| Treatment emergent SAE related to IMP as per Investigator's judgment | Primary SOC, HLGT, HLT and PT |
| TEAE leading to permanent intervention discontinuation | Primary SOC, HLGT, HLT and PT |
| | Primary SOC and PT |
| TEAE leading to death (death as an outcome of the AE as reported by the Investigator in the AE page) | Primary SOC, HLGT, HLT and PT |
| Pretreatment AE | Overview <sup>a</sup> |
| | Primary SOC and PT |

a Will include the following AE categories: any AEs, any serious AEs, any AEs leading to death, any AEs leading to permanent intervention discontinuation

## **Analysis of deaths**

In addition to the analyses of deaths included in Table 6 the number (%) of participants in the following categories will be provided:

- Deaths during the treatment-emergent and post-treatment periods
- Deaths in non-randomized or randomized but not treated participants

# Analysis of adverse events of special interest (AESIs) and other AEs of interest

Adverse events of special interest (AESIs) and other AEs of interest will be selected for analyses as indicated in Table 8. Number (%) of participants experiencing at least one event will be provided for each event of interest. Tables will be sorted as indicated in Table 6.

Table 8 - Selections for AESIs and other AEs of interest

| AE Grouping | Criteria |
|---|---|
| AESI | |
| Anaphylactic reaction | Anaphylactic reaction algorithmic approach (Introductory Guide for Standardised MedDRA Queries (SMQs) Version 18.1): includes anaphylactic reaction narrow SMQ (20000021) terms and programmatic identification of cases based on occurrence of at least two preferred terms meeting the algorithm criteria occurring within 24 hours of each other. The latter cases identified using the algorithm will undergo blinded medical review taking into account the timing of events relative to each other and to IMP administration for final determination of an anaphylactic reaction or not. |
| Systemic hypersensitivity reactions | SMQ [20000214] hypersensitivity narrow search and [AE corrective treatment/therapy='Y' or Action taken with IMP='Drug withdrawn' or Action taken with IMP='Drug interrupted'] followed by blinded medical review (documented process) for selection of relevant systemic hypersensitivity events |
| Helminthic infections | CMQ10544 based on HLGT as "Helminthic disorder" |
| Any severe type of conjunctivitis | CMQ10498 based on PTs (See Section 5.6) <sup>a</sup> and "Severe" ticked in Adverse Events eCRF page |
| Any severe type of blepharitis | CMQ10497 based on HLT as "Lid, lash and lacrimal infections, irritations and inflammations" and "Severe" ticked in Adverse Events eCRF page |
| Keratitis | CMQ10642 based on the following PTs [keratitis, allergic keratitis, ulcerative keratitis, atopic keratoconjunctivitis, herpes ophthalmic, ophthalmic herpes simplex, corneal infection] <sup>a</sup> |
| Clinically symptomatic eosinophilia (or eosinophilia associated with clinical symptoms) $\!\!^b$ | CMQ10641 based on HLT = Eosinophilic disorders or PT=Eosinophil count increased |
| Pregnancy of a female participants entered in a study as well as pregnancy occurring in a female partner of a male participant entered in a study with IMP/NIMP | "Pregnancy" or "Partner Pregnancy" checked on the<br>Pregnancy eCRF page as reported by the investigator |
| Significant ALT elevation | "ALT increase" and AESI answer "Yes" checked on AE eCRF as reported by the investigator (ALT >5 x ULN in participants with baseline ALT ≤2 x ULN; OR ALT >8 x ULN if baseline ALT >2 x ULN) |
| Symptomatic overdose with IMP | Symptomatic Overdose is answered Yes, with Overdose of IMP answered Yes on AE eCRF. |

| AE Grouping | Criteria |
|---|---|
| Symptomatic overdose with NIMP | Symptomatic Overdose is answered Yes, with Overdose of NIMP answered Yes on AE eCRF. |
| Other selected AE Grouping | |
| Serious injection site reactions or severe injection site reactions that last longer than 24 hours | HLT = 'Injection site reaction' and either with serious status, or with severe status and (AE end date/time - AE start date/time) ≥ 24 hours or ongoing |
| Severe or serious infection | Primary SOC = 'Infections and infestations' and with severe or serious status |
| Drug-related hepatic disorder | SMQ [20000006] Drug-related hepatic disorders- narrow |
| Injection site reaction | HLT = 'Injection site reaction' |
| Malignancy | SMQ [20000091] - Malignant or unspecified tumors narrow |
| Suicidal behavior | CMQ10639 based on the following PTs [Completed suicide, Suicidal ideation, Depression suicidal, Suicidal behavior, Suicide attempt] <sup>a</sup> |
| Conjunctivitis (narrow) | CMQ10644 based on the following PTs [Conjunctivitis, Conjunctivitis allergic, Conjunctivitis bacterial, Conjunctivitis viral, Atopic keratoconjunctivitis] <sup>a</sup> |
| Conjunctivitis (broad) | CMQ10645 based on the following PTs [Conjunctivitis, Conjunctivitis allergic, Conjunctivitis bacterial, Conjunctivitis viral, Atopic keratoconjunctivitis, Blepharitis, Dry eye, Eye irritation, Eye pruritus, Lacrimation increased, Eye discharge, Foreign body sensation in eyes, Photophobia, Xerophthalmia, Ocular hyperaemia, Conjunctival hyperaemia] <sup>a</sup> |
| Conjunctivitis (FDA) <sup>c</sup> | CMQ10643 based on the following PTs [Conjunctivitis, Conjunctivitis allergic, Conjunctivitis bacterial, Conjunctivitis viral, Eye irritation, Eye inflammation, Giant papillary conjunctivitis] <sup>a</sup> |
| Keratitis (FDA) <sup>C</sup> | CMQ30102 based on the following PTs in (keratitis, ulcerative keratitis, allergic keratitis, atopic keratoconjunctivitis, and ophthalmic herpes simplex) |

a The list of terms may be adjusted according to MedDRA version changes

## The following summaries will be provided:

- All TEAEs, by selected standardized MedDRA query (SMQ)/Customized MedDRA query (CMQ) and PT or by laboratory values (as in alanine aminotransferase (ALT) elevation), showing the number (%) of participants with at least 1 PT,
- For each AESI and other selected AE groupings,
  - Number (%) of participants with any specific TEAE

b All cases of Eosinophilia will be included in the analysis, where cases associated with clinical symptoms will be further described in the CSR

c FDA requested for US labeling

- Number (%) of participants with any specific serious AE (regardless of treatment emergent status)
- Number (%) of participants with any specific treatment emergent serious AE
- Number (%) of participants with any specific AE leading to death
- Number (%) of participants with any specific TEAE leading to permanent study drug discontinuation
- Number (%) of participants with any specific TEAE related to IMP reported by investigator
- Number (%) of participants with any specific TEAE by maximum intensity, corrective treatment, and final outcome
- Number of any specific TEAE adjusted by the exposure duration
- Number of participants with any specific TEAE adjusted by the exposure duration at risk. For each specific TEAE, Kaplan-Meier estimates of cumulative incidence at Week 12, and 24 and K-M plot may be provided to depict the course of onset over time if the number of events is large enough.
- Number (%) of participants with injection site reactions by IMP injection.
- Number (%) of participants with different number of injection site reactions.
- In addition, AESIs reported by the investigator in eCRF will be summarized separately.

In addition, the exposure-adjusted adverse event incidence rate tables will provide the number of patients with at least 1 event per 100 patient-years for the summaries of TEAEs, treatment emergent SAE, TEAE leading to permanent intervention discontinuation, and AESIs and other selected AE groups in Table 8

## 4.7.3 Additional safety assessments

#### 4.7.3.1 Laboratory variables, vital signs and electrocardiograms (ECGs)

The following laboratory variables, vital signs and electrocardiogram (ECG) variables will be analyzed. They will be converted into standard international units.

- Hematology:
  - Red blood cells and platelets and coagulation: hemoglobin, hematocrit, red blood cell count, platelet count
  - White blood cells: white blood cell count, neutrophils, lymphocytes, monocytes, basophils, eosinophils
- Clinical chemistry:
  - Metabolism: glucose, total cholesterol, total protein, creatine phosphokinase
  - Electrolytes: sodium, potassium, chloride, bicarbonate
- Renal function: creatinine, blood urea nitrogen, uric acid
- Liver function: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, lactate dehydrogenase, total bilirubin, albumin
- Pregnancy test: Serum β-human chorionic gonadotropin (all female participants) will be performed at screening (V1) in women of childbearing potential, and a urine pregnancy test will be performed at V2 and every 4 weeks thereafter.
- Hepatitis screen: hepatitis B surface antigen (HBs Ag), hepatitis B surface antibody (HBs Ab), hepatitis B core antibody (HBc Ab), hepatitis C virus antibodies (HCV Ab) will be tested at screening (V1). In case of results showing HBs Ag (negative) and HBc Ab (positive), an hepatitis B virus (HBV) deoxyribonucleic acid (DNA) testing will be performed and should be confirmed negative prior to randomization. In case of results showing HCV Ab (positive), an HCV ribonucleic acid (RNA) testing will be performed and should be confirmed negative prior to randomization.
- HIV screen: Anti-HIV-1 and HIV-2 antibodies will be tested at Visit 1.
- TB test (performed locally if required and results noted in the eCRF).

#### Urinalysis:

- Urinalysis will include specific gravity, pH, glucose, ketones, blood, protein, nitrate, leukocyte esterase, urobilinogen and bilirubin. If positive for protein and/or red blood cells, microscopic analysis will be performed by the central laboratory. Creatinine, leukotriene and tetranor PGDM will be tested by the central laboratory.
- Vital signs: pulse rate (beats per minute), systolic and diastolic blood pressure (mmHg) in a semi-supine or sitting position after 5 minutes, weight, respiratory rate (breaths per minute), temperature (degrees Celsius) and height (screening only).
- ECG variables: heart rate, PR, QRS, QT, and QTcF intervals after 10 minutes of rest in the supine position. Data are locally collected and read at screening (V1) and Week 24 (V6).

Data below the lower limit of quantitation/detection limit (LLOQ) will be replaced by half of the LLOQ, data above the upper limit of quantification will be replaced by ULOQ value.

#### Quantitative analyses

For all laboratory variables, vital signs and ECG variables above, descriptive statistics for results and changes from baseline will be provided for each analysis window, the last value and the worst value during the on-treatment period. These analyses will be performed using central measurements only (when available) for laboratory variables.

For all parameters, mean changes from baseline with the corresponding standard error will be plotted over time.

#### **Analyses according to PCSA**

Analysis of potentially clinically significant abnormality (PCSA) will be performed based on the PCSA list in effect at Sanofi at the time of the database lock. For parameters for which no PCSA criteria are defined, similar analyses will be done using the normal range, if applicable.

Analyses according to PCSA will be performed based on the worst value during the treatmentemergent period, using all measurements (either local or central, either scheduled, nonscheduled or repeated).

For laboratory variables, vital signs and ECG variables above, the incidence of participants with at least one PCSA during the treatment-emergent period will be summarized regardless of the baseline level and according to the following baseline status categories:

- Normal/missing
- Abnormal according to PCSA criterion or criteria

#### Additional analyses for suspect drug-induced liver injury

The following additional analyses will be performed for drug-induced liver injury:

- Time to onset of the initial ALT or aspartate aminotransferase (AST) elevation (>3 x ULN) and total bilirubin elevation (>2 x ULN) during the treatment-emergent period will be analyzed using Kaplan-Meier method.
- A graph of the distribution of peak values of ALT versus peak values of total bilirubin during the treatment-emergent period will be provided.
- For each liver function test (eg, ALT), participants having a PCSA (eg, ALT >5 ULN) will be summarized using the following categories: Returned to baseline PCSA status (or returned to value ≤ ULN in case of missing baseline) before last IMP dose, Returned to baseline PCSA status after last IMP dose, Never returned to baseline PCSA status, No assessment after elevation. This summary will be performed by categories of elevation (ALT >3, >5, >10, >20 ULN).

#### 4.8 OTHER ANALYSES

#### 4.8.1 Pharmacokinetic analyses

Predose dupilumab concentrations in serum at Visit 2 (Day 1), dupilumab trough concentrations at Week 4, Week 8, Week 12, Week 24/EOT Visit and post-treatment dupilumab concentrations at Week 36/EOS Visit will be provided.

Concentrations of dupilumab in serum will be summarized in the PK population using arithmetic and geometric means, SD, standard error of the mean (SEM), coefficient of variation (CV), minimum, median and maximum per sampling time. If date and/or time of the drug injection and/or sampling is missing then the concentration will not be taken into account. For drug-treated participants, where concentration values are below the lower limit of quantification (LLOQ),

one-half of the LLOQ will be used. Values will be expressed in the tables with no more than three significant figures. For participants in the placebo group, concentration values that are below the LLOQ will be taken into account with a plasma concentration considered equal to 0.

#### 4.8.2 Immunogenicity analyses

Anti-drug antibody (ADA) status to dupilumab (negative or titer value, if positive in the ADA assay) at Visit 2 (Day 1), Week 12, Week 24/EOT and follow up at Week 36 will be provided. The neutralizing antibody status for ADA positive samples will be provided.

Incidence will be provided for the following ADA response categories:

#### Pre-existing immunoreactivity is defined as:

An ADA positive response in the assay at baseline with all post first dose ADA results negative, OR an ADA positive response at baseline with all post first dose ADA responses less than 4-fold over baseline titer levels.

#### Treatment-emergent ADA response is defined as:

A positive response in the ADA assay post first dose, when baseline results are negative or missing.

# <u>Treatment-emergent ADA responses are further classified as Persistent, Indeterminate or Transient</u>

- a) Persistent Response- defined as a treatment-emergent ADA response with two or more consecutive ADA positive sampling time points, separated by greater than (>) 12-week period (84 days), with no ADA negative samples in between.
- b) Indeterminate Response- defined as a treatment-emergent response with only the last collected sample positive in the ADA assay
- c) Transient Response defined as a treatment-emergent response that is not considered persistent OR indeterminate

#### Treatment-boosted response is defined as:

An ADA positive response in the assay post first dose that is greater-than or equal to 4-fold over baseline titer levels, when baseline results are positive.

#### **Titer values** (Titer value category)

- Low (Titer < 1000)
- Moderate  $(1,000 \le \text{Titer} \le 10,000)$
- High (Titer >10,000)

The following summary will be provided based on ADA population:

- Number (%) of participants with pre-existing immunoreactivity
- Number (%) of participants with treatment-emergent ADA
- The summary statistics (including number, median, Q1, Q3, minimum and maximum) of the peak post-baseline titer for participants with treatment-emergent ADA, and participants with persistent, indeterminate and transient ADA response
- Number (%) of participant with transient treatment-emergent ADA
- Number (%) of participants with persistent treatment-emergent ADA
- Number (%) of participants with indeterminate treatment-emergent ADA
- Number (%) of participants with treatment-boosted ADA
- The summary statistics (including number, median, Q1, Q3, minimum and maximum) of the peak post-baseline titer for participants with treatment-boosted ADA
- The summary statistics (including number, mean, SD, median, Q1, Q3, minimum and maximum) of the ratio of peak post-baseline titer to baseline titer for participants with treatment-boosted ADA
- Listing of ADA peak titer levels and neutralizing antibody status
- Number (%) of participants with neutralizing antibody status

#### **Kinetics of treatment-emergent ADA response**

Number (%) of participants with treatment-emergent ADA positive response at each visit will be summarized, including titer categories (lower, moderate, and high titer), by each intervention group.

A plot of percentage of participants with treatment-emergent ADA positive response at each visit will be provided by each intervention group.

#### Association of Immunogenicity with Exposure, Safety and Efficacy

The safety and efficacy analyses mentioned below will be conducted using the following categories:

- ADA positive participants: Participants with treatment-emergent or treatment-boosted response.
- ADA negative participants: Participants with pre-existing immunoreactivity or negative in the ADA assay at all time points.

#### Association of ADA with PK

Associations between ADA variables (eg, ADA peak titers, neutralizing antibody status, treatment-emergent, persistent, indeterminate and transient response, treatment-boosted) and concentration of dupilumab in serum may be explored for each dupilumab dose group. A plot of

concentration of functional dupilumab versus visit will be provided by ADA classifications for the dupilumab dose group. Individual participant plots of dupilumab concentration according to ADA status will be provided to assess the impact of ADA on PK.

#### Association of ADA with clinical efficacy endpoints

Associations between the ADA variables (eg, ADA peak titers, neutralizing antibody status, treatment-emergent, persistent and treatment-boosted) and the primary efficacy endpoint may be explored for the dupilumab dosed group.

#### Association of ADA with clinical safety endpoints

Association of safety versus ADA status may be analyzed in the ADA population. The safety assessment may focus on the following events:

- Severe injection site reactions last longer than 24 hours or serious injection site reactions
- Hypersensitivity reactions (SMQ (20000214) hypersensitivity narrow search confirmed by medical review)
- Anaphylactic reactions (SMQ (20000021) anaphylactic reaction narrow search)

Associations between ADA variables (eg, ADA peak titers, neutralizing antibody status, treatment-emergent, persistent and treatment-boosted) and safety may be explored.

#### 4.8.3 Pharmacodynamic/genomics endpoints

Venous blood samples will be collected at Visit 2 (Week 0), Visit 3 (Week 4), Visit 4 (Week 8), Visit 5 (Week 12), Visit 6 (Week 24), and Visit 7 (Week 36), for measurement of total serum IgE. Total IgE will be measured using validated quantitative methods.

For those participants who consent to the optional pharmacogenetic/pharmacogenomic sample collection section of the ICF, blood (serum/plasma) for possible future analysis of potential biomarkers of drug response, disease activity, safety, and the type 2 inflammation pathway, and blood samples for exploratory genetic analysis of DNA or RNA will be collected and stored for possible future use. Participation is optional. Participants who do not wish to participate in the genetic research may still participate in the study.

Total IgE will be summarized in the safety population defined as participants who actually received at least 1 dose or part of a dose of the IMP. Baseline values will be the last value collected prior to the first IMP. Descriptive statistics (including number, mean, SD, median, Q1, Q3, min, max) of biomarkers at baseline will be summarized. In addition, for participants who take the prohibited medications/procedures or rescue medications defined in Table 5, the data after the medications will be censored and then last observation carried forward (LOCF) method will be implemented for missing data imputation in the analysis..

Summary plots (median with interquartile range) on values at each visit, absolute changes from baseline and percent changes from baseline will be provided for the total IgE by intervention group and visit.

Exploratory analysis of DNA, RNA and urine biomarkers will be addressed in a separate document.

#### 4.9 INTERIM ANALYSES

No interim analysis is planned.

A primary database lock will be performed when all randomized participants in this study have completed their 24-week treatment phase. Final analyses in the CSR will be based on this database.

The database will be updated at the end of the study for all participants to include the post-treatment follow-up information and updates for the events previously ongoing at the time of the primary lock. Additional data between this database lock and last participant completing last visit will be summarized in a CSR addendum.

#### 5 SUPPORTING DOCUMENTATION

#### 5.1 APPENDIX 1 LIST OF ABBREVIATIONS

ADA: anti-drug antibody
AE: adverse event

AESIs: adverse events of special interest

ALT: alanine aminotransferase ANCOVA: analysis of covariance AST: aspartate aminotransferase

ATC: anatomic category
CI: confidence interval
CLcr: creatinine clearance

CMH: Cochran-Mantel-Haenszel CMQ: customized MedDRA query

CSR: clinical study report

DLQI: Dermatology Life Quality Index

DNA: deoxyribonucleic acid ECG: electrocardiogram

eCRF: electronic case report form EMA: European Medicines Agency

EOT: end of treatment

EQ-5D-5L: 5-level EuroQol 5-dimensional questionnaire

FDA: Food and Drug Administration HADS: hospital anxiety and depression

HADS: hospital anxiety and depression scale HBc Ab: hepatitis B core antibody

HBs Ab: hepatitis B surface antibody
HBs Ag: hepatitis B surface antigen

HBV: hepatitis B virus

HCV Ab: hepatitis C virus antibodies HLGT: high level group term

HLT: high level term

HRQoL: health-related quality-of-life

IGA PN: Investigator's global assessment for prurigo nodularis

IMP: investigational medicinal product

ITT: intent-to-treat
LLT: lower-level term
LS: least squares

MedDRA: Medical Dictionary for Regulatory Activities PCSA: potentially clinically significant abnormality PGIC: Participant Global Impression of Change

PGIS: Global Impression of Severity

PK: pharmacokinetic PN: prurigo nodularis

Statistical Analysis Plan 08-Aug-2021 SAR231893 (REGN668) - EFC16460 - dupilumab Version number: 2

PT: preferred term
RNA: ribonucleic acid
SAE: serious adverse event
SAP: statistical analysis plan
SD: standard deviation

SDG: standardized drug grouping SMQ: standardized MedDRA query

SOC: system organ class

TEAE: treatment-emergent adverse event

ULN: upper limit of normal

WHO-DD: World Health Organization-Drug Dictionary

WI-NRS: worst-itch numeric rating scale WOCF: worst-observation carried forward

#### 5.2 APPENDIX 2 CHANGES TO PROTOCOL-PLANNED ANALYSES

This section summarizes major statistical changes in the protocol amendment.

Table 9 - Major statistical changes in protocol amendment(s)

| Amendment<br>Number | Approval<br>Date | Changes | Rationale |
|---|---|---|---|
| 1 | 20-May-2020 | To add "proportion of participants with Investigator's Global Assessment 0 or 1 score for PN-Stage (IGA PN-S) at Week 24" as another key secondary endpoint | To include a lesion-related key secondary endpoint according to the health authority's recommendations |
| | | To remove the endpoint "Change from baseline in PAS total score at Week 4, Week 8, Week 12, and Week 24" in the exploratory endpoint and modify the exploratory endpoint regarding the healed lesions from PAS questionnaire analysis | To clarify the analysis on efficacy evaluation of dupilumab on skin lesions using a modified prurigo activity score (PAS) 5-item questionnaire |
| | | To break out the secondary endpoints with multiple measuring timepoints into individual endpoints. | To clearly define the timepoints of each endpoint according to health authority's recommendation |
| | | To add the sensitivity analysis for secondary endpoints information, and to separate key secondary endpoints in a different row | To evaluate the robustness of the missing data imputation assumption by sensitivity analyses, and to clarify the endpoints analyses |
| | | To add the covariate "baseline anti-<br>depressant use (yes or no)" to primary and<br>secondary endpoint analyses | To adjust for potential impact of anti-<br>depressant use on the treatment effect<br>in primary and secondary efficacy<br>analyses |
| | | The following wording was added: "Data collected regarding the impact of the COVID-19 or other pandemics, on the participants will be summarized (eg, discontinuation due to COVID-19). Any additional analyses and methods required to investigate the impact of COVID-19 or other pandemics requiring public health emergency on the efficacy (eg, missing data due to COVID-19) and safety will be detailed in the SAP". | To describe alternative temporary mechanism that can be implemented in the study conduct in case of pandemic requiring public health emergency eg, COVID-19 |

### 5.3 APPENDIX 3 DEMOGRAPHICS AND BASELINE CHARACTERISTICS, PRIOR OR CONCOMITANT MEDICATIONS/PROCEDURES

#### Demographics, baseline characteristics, medical surgical history

The following demographics and baseline characteristics, medical and surgical history and disease characteristics at baseline will be summarized using descriptive statistics in the randomized population.

Demographic variables are

- Age in years (quantitative and qualitative variable: 18 40, 40 65, 65 75, and  $\ge 75$  years),
- Gender (Male, Female),
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or other Pacific Island, unknown),
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Unknown)
- Region (Asia: Taiwan, South Korea; East Europe: Hungary; Latin America: Chile; Western Countries: USA, Canada, France, Italy, Portugal, Spain, and UK)
- Territory (North America: USA, Canada; European Union: France, Italy, Portugal, Spain, Hungary, and UK; Rest of World: Taiwan, South Korea, Chile)
- Weight in kg (quantitative and qualitative variable:  $(<60, \ge 60 <90, \ge 90 \text{ kg})$
- BMI in kg/m<sup>2</sup> (quantitative and qualitative variable:  $<25, \ge 25 <30, \ge 30 \text{ kg/m}^2$ )

Baseline safety and efficacy parameters (apart from those listed above) will be presented along with the safety and efficacy summaries.

Medical (or surgical) history includes all the relevant medical (or surgical) history during the lifetime of the participant.

This information will be coded using the version of MedDRA currently in effect at Sanofi at the time of database lock.

Comorbidity will be summarized separately. The following comorbid diseases will be summarized from electronic case report form (eCRF) pages which were filled in by investigators based on participant reporting.

- Prurigo nodularis (Yes, Ongoing condition)
- Atopic dermatitis (Yes, Ongoing condition)
- Allergic rhinitis history (Yes, Ongoing condition)
- Allergic rhinoconjunctityitis (Yes, Ongoing condition)
- Asthma history (Yes, Ongoing condition)

- Food allergy history (Yes, Ongoing condition)
- Eosinophilic esophagitis history (Yes, Ongoing condition)

#### Disease characteristics at baseline

The following baseline disease characteristics will be summarized by intervention group:

- Duration of PN and grouping (years;  $\leq 3$  and  $\geq 3$ ) to be derived as
  - (Year of randomization Year of first diagnosis of PN) + (month of randomization month of first diagnosis of PN)/12
- Age of onset of PN (years)
- History of atopy (atopic or non-atopic)
  - Number of mild AD participants under atopic
- Stable use of TCS/TCI (yes or no)
- Baseline WI-NRS score
- Baseline IGA PN-S score (summary and frequency by each score level)
- Baseline IGA PN-A score (summary and frequency by each score level)
- Baseline skin Pain-NRS score
- Baseline Sleep-NRS score
- Baseline PGIS score
- PAS (number of prurigo lesions in a total and in representative area, and healed prurigo lesions) at baseline
- Baseline Hospital Anxiety and Depression Scale (HADS) total score
  - Baseline Hospital Anxiety score
  - Baseline Depression Scale score
- Baseline Dermatology Life Quality Index (DLQI) score
- Baseline EuroQol five dimensions questionnaire (ED-5D-5L) (single index score and VAS)
- Frequency of alcohol drinking in the past 12 months (never, occasional, at least monthly, at least weekly, at least daily) and number of drinks on a typical day (1 or 2, >2)
- Antidepressant use (yes or no) at baseline
- HIV (positive versus negative)

#### Prior or concomitant medications and procedure

All medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD) using the version currently in effect at Sanofi at the time of database lock.

All procedures will be coded to a PT and associated primary SOC using the version of MedDRA currently in effect at Sanofi at the time of database lock.

- Prior medications/procedures are those the participant used prior to first investigational medicinal product (IMP) injection. Prior medications/procedures can be discontinued before first administration or can be ongoing during treatment phase.
- Concomitant medications/procedures are any interventions received by the participant concomitantly to the IMP, from first administration of IMP to last IMP intake + 98 days.
- Post-treatment medications/procedures are those the participant took in the period running from the end of the concomitant medications period up to the end of the study.
- A given medication/procedure can be classified as a prior medication/procedure and/or as
  a concomitant medication/procedure and/or as post-treatment medication/procedure. If it
  cannot be determined whether a given medication/procedure was taken prior or
  concomitantly or post, it will be considered as prior, concomitant, and post-treatment
  medication/procedure.

The prior and concomitant medications/procedure will be summarized for the randomized population.

Medications will be summarized by intervention group according to the WHO-DD dictionary, considering the first digit of the anatomic category (ATC) class (anatomic category) and the first 3 digits of the ATC class (therapeutic category). All ATC codes corresponding to a medication will be summarized, and participants will be counted once in each ATC category (anatomic or therapeutic) linked to the medication. Therefore participants may be counted several time for the same medication.

The table for prior medications will be sorted by decreasing frequency of ATC followed by all other therapeutic classes based on the overall incidence across intervention groups. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

Concomitant medication received during first IMP to last IMP +14 days and concomitant medication received during first IMP to last IMP +98 days will be summarized separately. The tables for concomitant medications will be sorted by decreasing frequency of ATC followed by all other therapeutic classes based on the incidence in the dupilumab group. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

Medications will also be summarized by generic name sorted by decreasing frequency based on the incidence in the dupilumab group.

Procedures will be summarized by intervention group by primary SOC (sorted by internationally agreed order) and PT (sorted in alphabetical order), sorting is based on the overall incidence across intervention groups.

#### **Background** intervention

Participants will be required to apply moisturizers (emollients) once or twice daily for at least the 7 consecutive days immediately before baseline (Day 1) and continue until Week 36.

The compliance of moisturizers (emollients) used from 7 days before the baseline visit to Week 36 (or end of study), which is defined as the (number of days moisturizers used during the period) / (number of days within the period) x 100%, will be summarized by intervention group.

Similarly, the compliance of moisturizers (emollients) used from the baseline visit to Week 12 and Week 24 will be summarized by intervention group respectively.

In addition, the compliance of use of TCS/TCI from the baseline visit to Week 12 and Week 24 for participants with the stratification of stable use of TCS/TCI (yes) will be summarized by intervention group respectively.

.

#### Prohibited medications/procedures

The concomitant use of the following therapies is prohibited during the entire study. Study treatment will need to be discontinued in participants receiving these treatments:

- Systemic immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon gamma, Janus kinase inhibitors, azathioprine, methotrexate, hydroxychloroquine, dapsone, sulfasalazine, colchine, etc)
- Other monoclonal antibodies (which are biological modifiers)
- Phototherapy, including tanning beds
- Naltrexone or other opioid antagonist
- Gabapentin, pregabalin, and thalidomide

The concomitant use of the following therapies is prohibited except if the dose has been stable for at least 3 months prior to screening, but study treatment will not need to be discontinued in participants receiving the treatments listed below. The dose should also remain stable (can be reduced or discontinued if medically indicated) and should not be increased during the study.

- Paroxetine, fluvoxamine, or other SSRIs
- SNRIs
- Amitriptyline or other tricyclic or tetracyclic antidepressants

The concomitant use of the following therapies is also prohibited during the entire study, but study treatment will not need to be discontinued in participants receiving the treatments listed below:

• Intralesional corticosteroid injections and cryotherapy

- Sedating antihistamine
- Non-sedating antihistamine if used specifically for the treatment of itch secondary to AD or PN

The number and percentage of participants who take the prohibited medications/procedures will be provided. In addition, the time (week) of first prohibited medication/procedure taken will also be analyzed using Kaplan-Meier method.

#### Rescue medications

The following rescue medications may be used:

• Dermatological preparations of high potency or superpotent TCS and TCI.

If medically necessary (i.e., to control intolerable PN symptoms), rescue treatment for PN may be provided to study participants at the discretion of the Investigator.

Although the use of rescue medications is allowed at any time during the study, the use of rescue medications should be delayed, if possible, for at least 14 days following the initiation of the investigational treatment. The date and time of rescue medication administration as well as the name and dosage regimen of the rescue medication must be recorded in the eCRF.

• For the purpose of the efficacy responder analysis, a pre-specified algorithm will be used to classify rescue. In addition, a blinded review of all post-baseline medications to adjudicate rescue treatment, based on medical judgment, will be performed to adjudicate rescue. Participants who receive rescue treatment as per this adjudication during the study will be considered treatment failures.

The rescue medications will be analyzed by the same method as that used for prohibited medications/procedures.

#### 5.4 APPENDIX 4 DATA HANDLING CONVENTIONS

#### Demographic formulas

Age of onset of PN is calculated as:

Year of PN diagnosis – Year of birth

BMI is calculated as:

Weight in kg / (height<sup>2</sup> in meters)

#### **Renal function formulas**

For adults, creatinine clearance (CLcr) value will be derived using the equation of Cockroft and Gault:

CLcr (ml/min) = (140 - age) 
$$\times$$
 weight (kg)  $\times$  (1 - 0.15  $\times$  sex (0-M, 1-F))/ (0.814  $\times$  creatinine ( $\mu$ mol/l))

CLcr will be calculated using the last weight measurement on or before the visit of the creatinine measurement and age at the lab sampling day. Here age is calculated as following:

Age = age collected at screening + integer part of (lab sampling analysis day/365.25)

#### **Analysis windows for time points**

#### Efficacy assessment

For the efficacy assessment, the reference date for the derivation of relative days of events or findings will be the randomization day. If a participant receives IMP prior to the randomization by mistake, the reference date of efficacy assessment will be the date of the first IMP administration for that participant.

For daily eDiary data (WI-NRS, skin Pain-NRS, Sleep-NRS), all available values of daily measurements will be assigned to each week window according to Table 10, and then weekly average score will be calculated. Randomization day is used as the reference day (Day 1).

Table 10 - Time window for eDiary efficacy variables

| Time | Target day | Day range for calculating<br>weekly score |
|-------------------|------------|-------------------------------------------|
| Baseline (Week 0) | 1 | -7- <1 |
| Week 1 | 8 | 1-11 |
| Week 2 | 15 | 12-18 |
| Week 3 | 22 | 19-25 |
| Week 4 | 29 | 26-32 |
| Week 5 | 36 | 33-39 |
| Week 6 | 43 | 40-46 |
| Week 7 | 50 | 47-53 |
| Week 8 | 57 | 54-60 |
| Week 9 | 64 | 61-67 |
| Week 10 | 71 | 68-74 |
| Week 11 | 78 | 75-81 |

| Time | Target day | Day range for calculating weekly score |
|---------|------------|----------------------------------------|
| Week 12 | 85 | 82-88 |
| Week 13 | 92 | 89-95 |
| Week 14 | 99 | 96-102 |
| Week 15 | 106 | 103-109 |
| Week 16 | 113 | 110-116 |
| Week 17 | 120 | 117-123 |
| Week 18 | 127 | 124-130 |
| Week 19 | 134 | 131-137 |
| Week 20 | 141 | 138-144 |
| Week 21 | 148 | 145-151 |
| Week 22 | 155 | 152-158 |
| Week 23 | 162 | 159-165 |
| Week 24 | 169 | 166-172 |
| Week 25 | 176 | 173-179 |
| Week 26 | 183 | 180-186 |
| Week 27 | 190 | 187-193 |
| Week 28 | 197 | 194-200 |
| Week 29 | 204 | 201-207 |
| Week 30 | 211 | 208-214 |
| Week 31 | 218 | 215-221 |
| Week 32 | 225 | 222-228 |
| Week 33 | 232 | 229-235 |
| Week 34 | 239 | 236-242 |
| Week 35 | 246 | 243-249 |
| Week 36 | 253 | 250-256 |

For other efficacy variables, all available values of scheduled measurements will be assigned to the appropriate visit window according to Table 11. In the event of multiple measurements of the same test in the same window, the one closest to the targeted visit date will be used for the by-visit summary. If they are at the same number of days away from the target day, the latest one will be used.

08-Aug-2021 Version number: 2

Table 11 - Time window for efficacy variables

| | | Time windows for | | | | |
|---|---|---|---|---|---|---|
| Visit | Target<br>Day | DLQI,<br>IGA PN-A/PN-S | HADS,<br>EQ-5D-5L, Missed school/work<br>days | PGIS | PGIC | PAS |
| Visit 1 (Week -4 to -2) | <1 | | | <-14 | | <-14 |
| Visit 2 (Week 0) | 1 | 1- | 1- | -14-1 <sup>-</sup> | | -14-1- |
| Visit 3 (Week 4) | 29 | 1+-42 | | 1+-42 | 1+-42 | 1+-42 |
| Visit 4 (Week 8) | 57 | 43-70 | | 43-70 | 43-70 | 43-70 |
| Visit 5 (Week 12) | 85 | 71-126 | 1+-126 | 71-126 | 71-126 | 71-126 |
| Visit 6 (Week 24) | 169 | 127-210 | 127-210 | >126 | >126 | 127-210 |
| Visit 7 (Week 36) | 253 | >210 | >210 | | | >210 |

<sup>1-:</sup> up to randomization and before 1st dose date/time; 1+: after randomization or 1st dose date/time

#### Safety assessment

For the safety assessment, the reference date for the derivation of relative days of events or findings will be the date of first IMP administration. Selected safety variables will be summarized by the analysis window define in Table 12 for the by visit descriptive analysis. All available values from central lab will be assigned to the appropriate visit window. In the event of multiple measurements of the same test in the same window, the one closest to the targeted visit date will be used for the by-visit summary. If they are at the same number of days away from the target day, the latest one will be used. For procedures planned on Visit 2, if it is done on the same date as the first IMP injection but the performance time is missing, it will belong to Visit 2 time window.

Table 12 - Time window for safety endpoints

| | | | Time windows for | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Target Day | Vital signs | Hematology,<br>biochemistry | Urinalysis | CD4 T cell<br>count and<br>HIV test | Serum<br>Pregnancy<br>test | Urine Pregnancy<br>test | Physical examination | ECG |
| Visit 1 (Week -4<br>to -2) | <1 | <-14 | <-14 | <-14 | 1- | <-14 | | <-14 | 1- |
| Visit 2 (Week 0) | 1 | -14-1 <sup>-</sup> | -14-1 <sup>-</sup> | -14-1- | | | -14-1 <sup>-</sup> | -14-1 <sup>-</sup> | |
| Visit 3 (Week 4) | 29 | 1+-42 | 1+-42 | 1+-42 | | | 1+-42 | | |
| Visit 4 (Week 8) | 57 | 43-70 | 43-70 | 43-70 | | | 43-70 | | |
| Visit 5 (Week 12) | 85 | 71-126 | 71-126 | 71-126 | | | 71-126 | | |
| Visit 6 (Week 24) | 169 | 127-210 | 127-210 | >126 | 1+ | | 127-210 | 1+-210 | 1+ |
| Visit 7 (Week 36) | 253 | >210 | >210 | | | | >210 | >210 | |

<sup>1-:</sup> up to 1st dose date/time; 1+: after 1st dose date/time;

#### Pharmacokinetics/pharmacodynamics assessment

For the pharmacokinetics/pharmacodynamics variables summary, the reference date for the derivation of relative days of measurements will be the date of first IMP administration if the participant is treated with study treatment, or the randomization date if the participant is not treated. Pharmacokinetics /pharmacodynamics variables will be summarized by the analysis window defined in Table 13 for the by visit descriptive analyses. All available values of measurements will be assigned to the appropriate visit window. In the event of multiple measurements of the same test in the same window, the one closest to the targeted visit date will be used for the by-visit summary. If they are at the same distance to the target day, the latest one will be used. For procedures planned on Visit 2, if it is done on the same date as the first IMP injection but the performance time is missing, it will belong to Visit 2 time window.

Table 13 - Time window for pharmacokinetics/pharmacodynamics variables

| | | Time windows for | | |
|---|---|---|---|---|
| Visit | Target<br>day | Serum dupilumab concentration | Anti-drug antibodies | Total IgE |
| Visit 1 (Week -4) | <1 | | | |
| Visit 2 (Week 0) | 1 | 1- | 1 <sup>-</sup> | 1- |
| Visit 3 (Week 4) | 29 | 1+-42 | | 1+-42 |
| Visit 4 (Week 8) | 57 | 43-70 | | 43-70 |
| Visit 5 (Week 12) | 85 | 71-126 | 1⁺-126 | 71-126 |
| Visit 6 (Week 24) | 169 | 127-210 | 127-210 | 127-210 |
| Visit 7(Week 36) | 253 | >210 | >210 | >210 |

<sup>1-:</sup> up to 1st dose date/time or randomization if participant is not treated; 1+: after 1st dose date/time or randomization date if participant is not treated;

#### Unscheduled visits

Unscheduled visit measurements of laboratory data, vital signs, and ECG will be used for computation of baseline, the last on-treatment value, analysis according to PCSAs, and the shift summaries for safety. They will also be included in the by-visit summaries if they are re-allocated to scheduled visits.

#### 5.5 APPENDIX 5 SAMPLE SAS CODE

The multiple imputation and analysis model for the primary analysis of change from baseline in WI-NRS at Week 12 will be built with the following sample SAS code.

1. 40 datasets with a monotone missing pattern will be obtained, induced by Markov Chain Monte Carlo (MCMC) method on participants who have not taken the prohibited medications and/or rescue medications or have discontinued study treatment due to lack of efficacy prior to Week 12.

```
proc mi data=dat_etd seed=16460 nimpute=40 out=dat_mc;
    mcmc impute=monotone;
    var atopicyn stableyn region antidblyn trt01p winrsbl chg1winrs ...
    chg24winrs;
run;
```

2. For each of the imputed dataset with monotone missing pattern in step 1, the remaining missing data will be imputed using the regression method for the monotone pattern with adjustment for covariates including intervention groups, documented history of atopy (atopic or non-atopic), stable use of TCS/TCI (yes or no), region, baseline anti-depressant use (yes or no), and baseline value of the response variable.

```
proc mi data=dat_mc nimpute=1 seed=16461 out=dat_mi;
  by _imputation_;
  class atopicyn stableyn region antidblyn trt01p;
  monotone method=reg;
  var atopicyn stableyn region antidblyn trt01p winrsbl chg1winrs ...
  chg24winrs;
run;
```

3. Each of the 40 imputed datasets will be merged with the one dataset imputed by WOCF approach, and then be analyzed using the main statistical model. These 40 imputed datasets will be saved.

```
% w1
data dat imp;
     set dat mi wocf all;
Run;
proc sort data=dat imp;
     by _imputation_;
run;
proc glm data= dat imp;
     by _imputation ;
     class atopicyn stableyn region antidblyn trt01p;
     model chg24winrs = atopicyn stableyn region antidblyn
               trt01p winrsbl;
     lsmeans trt01p / stderr;
     estimate 'Diff Dupilumab vs Placebo' trt01p -1 1;
     ods output LSMeans=implsmeans Estimates=implsmeandiff;
run;
```

4. Applying Rubin's rule to combine analysis results (point estimates and standard errors) from 40 imputations using PROC MIANALYZE for the LS means and difference in LS means between dupilumab and placebo. Sample code:

```
proc sort data=implsMeans; by trt01pn _imputation_;run;
proc mianalyze data= implsmeans;
    by trt01pn;
    modeleffects lsmean;
    stderr stderr;
    ods output ParameterEstimates=lsmeans;
run;

proc mianalyze data=implsmeandiff;
    modeleffects estimate;
    stderr stderr;
    ods output ParameterEstimates=lsmeandiff;
run;
```

#### 5.6 APPENDIX 6 SELECTION CRITERIA FOR AE/MEDICATION GROUPINGS

Table 14 - List of PTs or Medications for CMQs/CDGs

| Grouping | Preferred Term/Medication Code | Preferred Term/Medication |
|---|---|---|
| Conjunctivitis | 10001257 | Adenoviral conjunctivitis |
| Conjunctivitis | 10010725 | Conjunctival irritation |
| Conjunctivitis | 10010726 | Conjunctival oedema |
| Conjunctivitis | 10010736 | Conjunctival ulcer |
| Conjunctivitis | 10010741 | Conjunctivitis |
| Conjunctivitis | 10010744 | Conjunctivitis allergic |
| Conjunctivitis | 10010745 | Conjunctivitis chlamydial |
| Conjunctivitis | 10010749 | Conjunctivitis gonococcal neonatal |
| Conjunctivitis | 10010754 | Conjunctivitis tuberculous |
| Conjunctivitis | 10010755 | Conjunctivitis viral |
| Conjunctivitis | 10018258 | Giant papillary conjunctivitis |
| Conjunctivitis | 10021629 | Inclusion conjunctivitis |
| Conjunctivitis | 10030861 | Ophthalmia neonatorum |
| Conjunctivitis | 10048908 | Seasonal allergy |
| Conjunctivitis | 10049458 | Herpes simplex virus conjunctivitis neonatal |
| Conjunctivitis | 10051625 | Conjunctival hyperaemia |
| Conjunctivitis | 10053991 | Inclusion conjunctivitis neonatal |
| Conjunctivitis | 10061784 | Conjunctivitis bacterial |
| Conjunctivitis | 10062889 | Pingueculitis |
| Conjunctivitis | 10063669 | Photoelectric conjunctivitis |
| Conjunctivitis | 10067317 | Oculorespiratory syndrome |
| Conjunctivitis | 10067817 | Acute haemorrhagic conjunctivitis |
| Conjunctivitis | 10069166 | Blebitis |
| Conjunctivitis | 10071570 | Ligneous conjunctivitis |
| Conjunctivitis | 10074701 | Noninfective conjunctivitis |
| Conjunctivitis | 10075264 | Oculoglandular syndrome |
| Conjunctivitis | 10080825 | Conjunctivitis fungal |
| Conjunctivitis | 10084034 | Conjunctival suffusion |
| Intravenous immunoglobulin therapy | CAS 8000012671 | IMMUNOGLOBULIN HUMAN NORM |
| Intravenous immunoglobulin therapy | CAS 8000050682 | IMMUNOGLOBULIN, PORCINE |
| Intravenous immunoglobulin therapy | CAS 8000056919 | IMMUNOGLOBULIN G HUMAN |

| Grouping | Preferred Term/Medication Code | Preferred Term/Medication |
|---|---|---|
| Intravenous immunoglobulin therapy | CAS 8600000563 | IMMUNOGLOBULINS NOS |
| Intravenous immunoglobulin therapy | CAS 8600001670 | IMMUNOGLOBULIN HUMAN NORMAL<br>SLRA |
| Intravenous immunoglobulin therapy | CAS 8600001671 | IMMUNOGLOBULIN HUMAN NORMAL<br>IFAS |
| Intravenous immunoglobulin therapy | RECNO 900708 | OTHER IMMUNOGLOBULINS |
| Intravenous immunoglobulin therapy | RECNO 900722 | IMMUNE SERA AND IMMUNOGLOBULINS |
| Intravenous immunoglobulin therapy | RECNO 900728 | IMMUNOGLOBULINS |
| Intravenous immunoglobulin therapy | RECNO 900914 | SPECIFIC IMMUNOGLOBULINS |
| Intravenous immunoglobulin therapy | RECNO 901112 | IMMUNOGLOBULINS, NORMAL<br>HUMAN |

Abbreviations: CAS: Chemical Abstract Service Registry Number RECNO: Drug Record Number

#### 5.7 APPENDIX 7 MEDICATION/PROCEDURE ADJUDICATION ALGORITHM

Algorithm for determining whether treatment with following medications or procedures constitutes treatment failure resulting in setting data as non-responder after taking medication or undergoing procedure in the main statistical analysis

- 1. Not required to adjudicate post-baseline medications (WHODD-coded) or procedures (CMQ-coded) as these will be considered treatment failures if used at any time<sup>1</sup>.
  - a) Always considered treatment failure
    - ATC2 = CORTICOSTEROIDS FOR SYSTEMIC USE
    - ATC2 = IMMUNOSUPPRESSANTS (systemic, e.g. oral or parenteral route)
    - Preferred Drug Name = Ciclosporin
    - Preferred Drug Name = Methotrexate
    - Preferred Drug Name = Mycophenolate sodium
    - Preferred Drug Name = Mycophenolic acid
    - Preferred Drug Name = Azathioprine
    - Preferred Drug Name = Gabapentin
    - Preferred Drug Name = Pregabalin
    - Preferred Drug Name = Thalidomide
    - Preferred Drug Name = Lenalidomide
    - Preferred Drug Name = Baricitinib
    - Preferred Drug Name = Ruxolitinib
    - Preferred Drug Name = Tofacitinib
    - Preferred Drug Name = AbrocitinibPreferred Drug Name = Delgocitinib
    - Preferred Drug Name = Nalbuphine
    - Preferred Drug Name = Naltrexone
    - Preferred Drug Name = Naloxone
    - Preferred Drug Name = Vixarelimab
    - Preferred Drug Name = Nemolizumab
    - Preferred Drug Name = Serlopitant
    - Preferred Drug Name = Aprepitant
    - CMQb HLT Phototherapies
    - CMQ Tanning single PT

- b) Never considered treatment failure:
  - ATC2 = EMOLLIENTS AND PROTECTIVES
  - ATC2 = GENERAL NUTRIENTS
  - ATC2 = VITAMINS
  - ATC2 = ANTIVIRALS FOR SYSTEMIC USE
  - ATC2 = ANTIFUNGALS FOR DERMATOLOGICAL USE
  - ATC2 = ANTISEPTICS AND DISINFECTANTS
  - ATC2 = ANTIBIOTICS AND CHEMOTHERAPEUTICS FOR DERMATOLOGICAL USE
  - ATC2 = ANTI-ACNE PREPARATIONS, excluding D10AA Corticosteroids, combinations for treatment of acne
  - ATC2 = OPHTHALMOLOGICALS
  - ATC1 = ANTIINFECTIVES FOR SYSTEMIC USE, excluding D07C Corticosteroids, combinations with antibiotics
  - ATC1 = BLOOD AND BLOOD FORMING ORGANS
  - ATC1 = ALIMENTARY TRACT AND METABOLISM
  - ATC1 = MUSCULO-SKELETAL SYSTEM, excluding M01BA Antiinflammatory/antirheumatic agents in combination with corticosteroids
  - ATC2 = COUGH AND COLD PREPARATIONS
  - ATC2= PSYCHOLEPTICS, excluding N05BB Diphenylmethane derivatives and N05C HYPNOTICS AND SEDATIVES

<sup>1</sup> A blinded review of all post-baseline medications or procedures to adjudicate whether treatment constitutes treatment failure, based on medical judgment, may be performed in addition. A listing of treatments or procedures classified as treatment failure in a manner inconsistent with the classification under #1 will be provided, along with supporting rationale.

## 2. Require to adjudicate medications or procedures that may constitute treatment failure

- All other medications and procedures listed in the protocol and Table 5 of the SAP (not noted in 1. above) given for indications consistent with PN<sup>2</sup>
- Considerations in determining treatment failure include the criteria already set forth in Table 5 of the SAP in addition to the type of medication or procedure, indication, dose, route of administration, timing, frequency and the potential impact of the use of the prohibited medications/procedures and rescue medications on the primary and key secondary efficacy endpoints.
- 2 Below is a list of indications consistent with PN based on PT level from concomitant medication/procedure data using MedDRA dictionary

| System Organ Class | High Level Term | Preferred Term | Preferred Term Code |
|---|---|---|---|
| Skin and subcutaneous tissue disorders | Dermatitis and eczema | Neurodermatitis | 10029263 |
| Infections and infestations | Bacterial infections NEC | Eczema impetiginous | 10051890 |
| Infections and infestations | Skin structures and soft tissue infections | Dermatitis infected | 10012470 |
| Infections and infestations | Skin structures and soft tissue infections | Eczema infected | 10014199 |
| Skin and subcutaneous tissue disorders | Dermatitis and eczema | Dermatitis | 10012431 |
| Skin and subcutaneous tissue disorders | Dermatitis and eczema | Dermatitis atopic | 10012438 |
| Skin and subcutaneous tissue disorders | Dermatitis and eczema | Eczema | 10014184 |

#### 6 REFERENCES

1. Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71.

# Signature Page for VV-CLIN-0602730 v2.0 efc16460-16-1-9-sap

| Approve & eSign |
|-----------------|
| Approve & eSign |